Protocol Title: Evaluation of Daily Disposable Silicone Hydrogel Multifocal Toric Contact

Lenses

Protocol Number: CR-6435

Version: 1.0

Date: 12 May 2021

Test Articles: JJVC Investigational Multifocal Toric Contact Lenses manufactured in

Senofilcon A (C3) material with UV/HEV blocker

Key Words: Presbyopia, Multifocal, Astigmatism, Daily Wear, Daily Disposable,

Dispensing, senofilcon A, logMAR visual acuity, CLUE questionnaire

#### Statement of Compliance to protocol, GCP and applicable regulatory guidelines:

This trial will be conducted in compliance with the protocol, ISO 14155,<sup>1</sup> the International Conference on Harmonization Good Clinical Practice E6 (ICH-GCP),<sup>2</sup> the Declaration of Helsinki,<sup>3</sup> and all applicable regulatory requirements.

#### **Confidentiality Statement:**

This document contains confidential information, which should not be copied, referred to, released or published without written approval from Johnson & Johnson Vision Care, Inc. The information may not be disclosed to others except to the extent necessary to obtain Institutional Review Board/Independent Ethics Committee approval and informed consent, or as required by International, Federal and State Laws, as applicable. Persons to whom this information is disclosed must be informed that this information is privileged and confidential and that it should not be further disclosed without the written permission of Johnson & Johnson Vision Care, Inc. Any supplemental information that may be added to this document is also confidential and proprietary to Johnson & Johnson Vision Care, Inc. and must be kept in confidence in the same manner as the contents of this document.

| TABLI | E OF CONTENTS | |
|---|---|---|
| PROTO | OCOL TITLE, NUMBER, VERSION AND DATE | 6 |
| <b>SPONS</b> | OR NAME AND ADDRESS | 6 |
| <b>MEDIC</b> | CAL MONITOR | 6 |
| | ORIZED SIGNATURES | |
| CHANG | GE HISTORY | 9 |
| SYNOF | PSIS | 10 |
| COMM | IONLY USED ABBREVIATIONS, ACRONYMS AND DEFINITIONS OF TER | RMS |
| | ······································ | |
| 1. IN | TRODUCTION AND BACKGROUND | |
| 1.1. | Name and Descriptions of Investigational Products | 18 |
| 1.2. | Intended Use of Investigational Products | |
| 1.3. | Summary of Findings from Nonclinical Studies | 18 |
| 1.4. | Summary of Known Risks and Benefits to Human Subjects | |
| 1.5. | Relevant Literature References and Prior Clinical Data Relevant to Proposed Clin | nica |
| Study | y | 18 |
| 2. ST | UDY OBJECTIVES, ENDPOINTS AND HYPOTHESES | 19 |
| 2.1. | Objectives | 19 |
| 2.2. | Endpoints | 19 |
| 2.3. | Hypotheses | 20 |
| 3. TA | ARGETED STUDY POPULATION | 21 |
| 3.1. | General Characteristics | 21 |
| 3.2. | Inclusion Criteria | 21 |
| 3.3. | Exclusion Criteria | 22 |
| 3.4. | Enrollment Strategy | 23 |
| 4. ST | UDY DESIGN AND RATIONALE | 23 |
| 4.1. | Description of Study Design | 23 |
| 4.2. | Study Design Rationale | 23 |
| 4.3. | Enrollment Target and Study Duration | |
| 5. TE | EST ARTICLE ALLOCATION AND MASKING | 24 |
| 5.1. | Test Article Allocation | 24 |
| 5.2. | Masking | |
| 5.3. | Procedures for Maintaining and Breaking the Masking | |
| 6. ST | UDY INTERVENTION | 25 |
| 6.1. | Identity of Test Articles | 25 |
| 6.2. | Ancillary Supplies/Products | 26 |
| 6.3. | Administration of Test Articles | 26 |
| 6.4. | Packaging and Labeling | |
| 6.5. | Storage Conditions | 27 |
| 6.6. | Collection and Storage of Samples | |
| 6.7. | Accountability of Test Articles | 27 |
| 7. ST | UDY EVALUATIONS | |
| 7.1. | Time and Event Schedule. | |
| 7.2. | Detailed Study Procedures | 29 |
| VI | SIT 1 | 20 |

| VISI | TT 2 | 37 |
|--------|----------------------------------------------------------|----|
| VISI | TT 3 | 43 |
| VISI | T 4 | 47 |
| FINA | AL EVALUATION | 49 |
| 7.3. | Unscheduled Visits | 50 |
| 7.4. | Laboratory Procedures | 52 |
| 8. SUB | JECTS COMPLETION/WITHDRAWAL | 52 |
| 8.1. | Completion Criteria | 52 |
| 8.2. | Withdrawal/Discontinuation from the Study | 52 |
| 9. PRE | -STUDY AND CONCOMITANT INTERVENTION/MEDICATION | 53 |
| 9.1. | Systemic Medications | 53 |
| 10. DE | EVIATIONS FROM THE PROTOCOL | 54 |
| 11. ST | UDY TERMINATION | 55 |
| 12. PR | COCEDURE FOR HANDLING PRODUCT QUALITY COMPLAINTS | 56 |
| 13. AI | OVERSE EVENTS | |
| 13.1. | Definitions and Classifications | 57 |
| 13.2. | Assessing Adverse Events | 59 |
| 13.2 | .1. Causality Assessment | 59 |
| _ | .2. Severity Assessment | 60 |
| 13.3. | Documentation and Follow-Up of Adverse Events | 60 |
| 13.4. | Reporting Adverse Events | 61 |
| 13.4 | 1 0 | |
| 13.4 | | |
| 13.5. | Event of Special Interest | |
| 13.6. | Reporting of Pregnancy | |
| | ATISTICAL METHODS | |
| 14.1. | General Considerations | |
| 14.2. | Sample Size Justification | |
| 14.3. | Analysis Populations | |
| 14.4. | Level of Statistical Significance | |
| 14.5. | Primary Analysis | |
| 14.6. | Secondary Analysis | |
| 14.7. | Other Exploratory Analyses | |
| 14.8. | Interim Analysis | |
| 14.9. | Procedure for Handling Missing Data and Drop-Outs | |
| 14.10. | Procedure for Reporting Deviations from Statistical Plan | |
| | ATA HANDLING AND RECORD KEEPING/ARCHIVING | |
| 15.1. | Electronic Case Report Form/Data Collection | |
| 15.2. | Subject Record | |
| 15.3. | Trial Registration on ClinicalTrials.gov | |
| _ | ATA MANAGEMENT | |
| 16.1. | Access to Source Data/Document | |
| 16.2. | Confidentiality of Information | |
| 16.3. | Data Quality Assurance | |
| 16.4. | Data Monitoring Committee (DMC) | 72 |

| 17. CLINICAL MONITORING | 72 |
|---|---|
| 18. ETHICAL AND REGULATORY ASPECTS | |
| 18.1. Study-Specific Design Considerations | |
| 18.2. Investigator Responsibility | |
| 18.3. Independent Ethics Committee or Institutional Review Board (IEC/IRB) | |
| 18.4. Informed Consent | |
| 18.5. Privacy of Personal Data | |
| 19. STUDY RECORD RETENTION | |
| 20. FINANCIAL CONSIDERATIONS | |
| 21. PUBLICATION | |
| 22. REFERENCES | |
| APPENDIX A: PATIENT REPORTED OUTCOMES (STUDY QUESTIONNAIRES | |
| APPENDIX B: PATIENT INSTRUCTION GUIDE | |
| APPENDIX C: PACKAGE INSERT (APPROVED PRODUCT) | |
| APPENDIX D: LENS FITTING GUIDE | |
| APPENDIX E: PRESBYOPIC SYMPTOMS QUESTIONNAIRE | |
| APPENDIX F: OCULAR DOMINANCE | |
| APPENDIX G: BINOCULAR OVER REFRACTION | |
| APPENDIX H: DETERMINATION OF NEAR ADDITION | 111 |
| NEAR LOGMAR VISUAL ACUITY MEASUREMENT PROCEDURE | |
| LENS FITTING CHARACTERISTICS | |
| SUBJECT REPORTED OCULAR SYMPTOMS | 126 |
| DETERMINATION OF DISTANCE SPHEROCYLINDRICAL REFRAC | TIONS |
| | 128 |
| BIOMICROSCOPY SCALE | 134 |
| KERATOMETRY | |
| DISTANCE AND NEAR VISUAL ACUITY EVALUATION | 142 |
| TORIC FIT EVALUATION | |
| DISTANCE LOGMAR VISUAL ACUITY MESAUREMENT PROCE | EDURE |
| VISUAL ACUITY CHART LUMINANCE AND ROOM ILLUMINA | ATION |
| TESTING | |
| APPENDIX I: GUIDELINES FOR COVID-19 RISK MITIGATION | |
| PROTOCOL COMPLIANCE INVESTIGATOR(S) SIGNATURE PAGE | 177 |
| LIST OF FIGURES | |
| Figure 1: Study Flowchart | 15 |
| rigule 1. Study Flowchaft | 13 |
| LIST OF TABLES | |
| Table 1: Test Articles | 25 |
| Table 2: Ancillary Supplies | |
| Table 3: Time and Events | |
| Table 4: Disallowed systemic medications | |
| Table 5: Examples of major and minor protocol deviations | |

| Table 6: Historical Binocular High Luminance High Contrast Visual Performance | 64 |
|---|---|
| Table 7: Historical CLUE Scores – 2-Week Follow-up | 64 |
| Table 8: Sample Size Estimates for Primary Endpoints | 65 |
| Table 9: Power Analysis for Secondary Endpoints | 65 |

#### PROTOCOL TITLE, NUMBER, VERSION AND DATE

Protocol Title: Evaluation of Daily Disposable Silicone Hydrogel Multifocal Toric Contact

Lenses

Protocol Number: CR-6435

Version: 1.0

Date: 12 May 2021

#### **SPONSOR NAME AND ADDRESS**

Johnson & Johnson Vision Care (JJVC) 7500 Centurion Parkway Jacksonville, FL 32256

# MEDICAL MONITOR

The Medical Monitor must be notified by the clinical institution/site by e-mail, fax, or telephone within 24 hours of learning of a Serious Adverse Event. The Medical Monitor may be contacted during business hours for adverse event questions. General study related questions should be directed towards your assigned clinical research associate.

The Medical Monitoring Plan is maintained as a separate document and included in the Trial Master File.

#### **AUTHORIZED SIGNATURES**

The signatures below constitutes the approval of this protocol and the attachments and provide the necessary assurances that this trial will be conducted according to all stipulations of the protocol, including all statements regarding confidentiality, and according to local legal and regulatory requirements and applicable U.S. federal regulations,<sup>4</sup> ICH guidelines,<sup>2</sup> ISO 14155,<sup>1</sup> and the Declaration of Helsinki.<sup>3</sup>

| Author | See Electronic Signature Page | |
|--------------------------------|-------------------------------|------|
| | | DATE |
| Clinical Operations<br>Manager | See Electronic Signature Page | |
| J | | DATE |
| Biostatistician | See Electronic Signature Page | |
| | | DATE |
| Biostatistics<br>Reviewer | Saa Elaatrania Signatura Daga | |
| Reviewei | See Electronic Signature Page | DATE |
| Data Management | See Electronic Signature Page | DATE |
| | | DAIL |
| Medical Safety | | |
| Officer | See Electronic Signature Page | DATE |

| Reviewer | See Electronic Signature Page | |
|----------|-------------------------------|------|
| | | DATE |
| Approver | See Electronic Signature Page | |
| | | DATE |

## **CHANGE HISTORY**

| Version | Originator | Description of Change(s) and Section | Date |
|---------|------------|--------------------------------------|-------------|
| | | Number(s) Affected | |
| 1.0 | | Original Protocol | 12 May 2021 |

## **SYNOPSIS**

| Protocol Title | Evaluation of Daily Disposable Silicone Hydrogel Multifocal |
|---|---|
| C | Toric Contact Lenses |
| Sponsor | JJVC, 7500 Centurion Parkway, Jacksonville, FL 32256 |
| Clinical Phase | Clinical trial phase: Confirmatory |
| T: 1D : : : | Design control phase: 2b |
| Trial Registration | This study will be registered on ClinicalTrials.gov based on<br>the following: The purpose of the study is for design<br>confirmation, not feasibility. |
| Test Article | Investigational Products: JJVC Investigational Multifocal |
| | Toric Contact Lenses manufactured in Senofilcon A (C3) material with UV/HEV blocker |
| Wear and Replacement<br>Schedules | Wear Schedule: The lenses will be used on a daily disposable basis. |
| | Replacement Schedule: The lenses will be replaced each day of wear or if lost or damaged. |
| Objectives | The purpose of the study is to confirm the performance of the study lens relative to previously established safety and efficacy criteria. Study results may also be compared to the results obtained in other studies through aggregation of results in graphs and tables. |
| | Primary Objective The primary objectives of this study are to assess the clinical performance of investigational multifocal toric contact lenses with respect to subjective vision measured via CLUE <sup>TM</sup> questionnaire, and visual acuity (logMAR) after approximately two weeks of lens wear. |
| | Secondary Objective The secondary objectives of this study are to compare the clinical performance of investigational multifocal toric contact lenses with the subjects' habitual correction with respect to subjective vision, comfort and lens handling measured via the CLUE <sup>TM</sup> questionnaire after approximately two weeks of lens wear. |
| | Exploratory Objectives Additional exploratory objectives are to evaluate the lens fit acceptance and toric fit of the investigational multifocal toric lenses, and the ocular health via slit lamp findings. |

| Study Endpoints | All secondary and primary endpoints are considered at the 2- |
|---|---|
| Study Enapoints | week follow-up in the optimized lenses (Visit 4). |
| | Primary endpoints: • Binocular high luminance, high contrast logMAR visual acuity at distance (4 m), intermediate (64 cm), and near (40 cm) at 2-week follow-up |
| | • Subjective vision via CLUE <sup>TM</sup> questionnaire at 2-week follow-up |
| | Secondary endpoints: • Subjective vision score via CLUE <sup>TM</sup> questionnaire: change from baseline to 2-week follow-up |
| | • Subjective comfort score via CLUE™ questionnaire: change from baseline to 2-week follow-up |
| | Subjective handling score via CLUE <sup>TM</sup> questionnaire: change from baseline to 2-week follow-up |
| | Exploratory endpoints: • Percentage of eyes with an unacceptable lens fit during the study |
| | • Percentage of lens fits with rotation stability within 5 degrees at 15 minutes after insertion at the fitting visit |
| | • Percentage of lens fits with absolute rotation error within 10 degrees at 15 minutes after insertion at the fitting visit |
| | Percentage of eyes with Grade 3 or 4 findings during the post-fit period. |
| Study Design | The study is a bilateral, single-masked, single-arm, 4-visit dispensing study. There will be one study treatment, with the subject being dispensed lenses for 6 to 8 days, then will return for lens optimization (if needed). Following the optimization visit, the study lenses will be worn for approximately two |
| | weeks, including a follow-up visit after 6 to 8 days. The primary endpoints will be logMAR visual acuity at distance, intermediate and near and subjective vision scores. See the flow chart at the end of the synopsis table for the schematic of the study visits and procedures of main |
| | observations. |

| Commis Size | Ammovimotoly, 50 myonia sylvinta syvida assissa 411- |
|---|---|
| Sample Size | Approximately 50 myopic subjects with against-the-rule astigmatism will be enrolled, with the aim that at least 45 will complete the study. Approximately 40 hyperopic subjects with against-the-rule astigmatism will be enrolled, with the aim that at least 35 will complete the study. The study lenses for the hyperopic subjects are likely to be available before the |
| | lenses for the myopic subjects, therefore, the study may enroll and complete all hyperopes before myopes are enrolled. |
| Study Duration | Lenses in minus powers and plus powers will be evaluated in two separate phases of the study which may run at different times depending on when lenses become available. Each |
| | phase of the study will last approximately 3 months. Each individual subject is expected to be in the study for approximately 3 weeks. |
| Anticipated Study<br>Population | Healthy male and female volunteers with presbyopia, ametropia (hyperopia or myopia) and astigmatism will be screened as per criteria outlined below. All volunteers will have baseline measurements taken to ensure eligibility. The baseline procedures will occur after informed consent has been obtained. For a detailed list of procedures see the time and events schedule listed below. |
| Eligibility Criteria -<br>Inclusion | Potential subjects must satisfy all of the following criteria to be enrolled in the study: |
| | Inclusion Criteria following Screening The subject must: |
| | <ol> <li>Read, understand, and sign the STATEMENT OF<br/>INFORMED CONSENT and receive a fully executed<br/>copy of the form.</li> <li>Appear able and willing to adhere to the instructions</li> </ol> |
| | set forth in this clinical protocol. 3. Be at least 40 and not more than 70 years of age at the time of screening. |
| | 4. Own a wearable pair of spectacles if required for their distance vision. |
| | 5. Be an adapted soft contact lens wearer in both eyes (i.e. worn lenses for at least 8 hours per day at least two days per week for the past 4 weeks). |
| | 6. Be already wearing a presbyopic contact lens correction (e.g., reading spectacles over contact lenses, multifocal or monovision contact lenses, etc.) or if not respond positively to at least one symptom on the "Presbyopic Symptoms Questionnaire". |

| | _ |
|---|---|
| | Inclusion Criteria at Baseline Evaluation: |
| | <ol> <li>7. The subject's distance spherical component of their refraction must be in the range of either -1.25 D to -3.75 D, or +1.25 D to +3.75 D.</li> <li>8. The subject's refractive cylinder must be -1.00 D to -1.50 D in each eye, with the cylinder axes in the range of 90°±30°.</li> <li>9. The subject's ADD power must be in the range of +0.75 D to +2.50 D in each eye.</li> <li>10. The subject must have best corrected distance visual acuity of 20/20-3 or better in each eye.</li> </ol> |
| Eligibility Criteria - | Potential subjects who meet any of the following criteria will |
| Exclusion | be excluded from participating in the study: |
| | Exclusion Criteria following Screening |
| | The subject must not: |
| | The subject must not. |
| | <ol> <li>Be currently pregnant or lactating.</li> <li>By self-report, have any systemic disease (e.g. Sjögren's Syndrome), allergies, infectious disease (e.g., hepatitis, tuberculosis), contagious immunosuppressive diseases (e.g., HIV), autoimmune disease (e.g. rheumatoid arthritis), or other diseases, by self-report, which are known to interfere with contact lens wear and/or participation in the study.</li> <li>Use systemic medications that may interfere with contact lens wear or cause blurred vision. See Section 9.1 for additional details regarding excluded systemic medications.</li> <li>Currently use ocular medication (with the exception of rewetting drops).</li> <li>Have any known hypersensitivity or allergic reaction to single use preservative free rewetting drops or sodium fluorescein.</li> <li>Have had any previous, or have any planned, ocular or intraocular surgery (e.g. radial keratotomy, PRK, LASIK,</li> </ol> |
| | <ul> <li>cataract surgery, retinal surgery, etc.).</li> <li>7. Have had previous eyelid injuries, surgeries or procedures which are known to have caused abnormal eyelid position or movement, by self-report.</li> <li>8. Have participated in any contact lens or lens care product</li> </ul> |
| | clinical trial within 7 days prior to study enrollment. |

| | <ul> <li>9. Be an employee or immediate family member of an employee of clinical site (e.g., Investigator, Coordinator, Technician).</li> <li>10. Have a history of amblyopia or strabismus, by self-report.</li> <li>11. Have a history of herpetic keratitis, by self-report.</li> </ul> |
|---|---|
| | Exclusion Criteria at Baseline Evaluation The subject must not: |
| | <ul> <li>12. Have ocular allergies, infections or other ocular abnormalities that are known to interfere with contact lens wear and/or participation in the study. This may include, but not be limited to entropion, ectropion, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions, aphakia, or corneal distortion</li> <li>13. Have any Grade 3 or greater slit lamp findings (e.g., edema, corneal neovascularization, corneal staining, tarsal abnormalities, conjunctival injection) on the FDA scale.</li> </ul> |
| Disallowed<br>Medications/Interventions | Use of any prescription or over-the-counter (OTC) medications that may affect contact lens wear. See Section 9.1 for details regarding disallowed systemic medications. |
| Measurements and Procedures | logMAR visual acuity and subjective responses for vision, comfort and lens handling using the CLUE questionnaire. |
| Microbiology or Other<br>Laboratory Testing | None |
| Study Termination | The occurrence of one or more Unanticipated Adverse Device Effect (UADE), or any SAE where relationship to study agent cannot be ruled out, may result in stopping the further dispensing of investigational product. In the event of a UADE or SAE, the Sponsor Medical Monitor may unmask the treatment regimen of subject(s) and may discuss this with the Principal Investigator before any further subjects are enrolled. |
| Ancillary Supplies/ Study-<br>Specific Materials | Rewetting drops and saline for storing worn lenses. Lens vials and caps and materials for returning worn contact lenses will be supplied to sites. |
| Principal Investigator(s) and Study Institution(s)/Site(s) | A full list of Principal Investigators, clinical sites, and institutions is kept separately from the Study Protocol and is included in the study Trial Master File. |

Figure 1: Study Flowchart



# COMMONLY USED ABBREVIATIONS, ACRONYMS AND DEFINITIONS OF TERMS

ADD Plus Power Required For Near Use

ADE Adverse Device Effect

AE Adverse Event/Adverse Experience
BCVA Best Corrected Visual Acuity

BSCVA Best Spectacle Corrected Visual Acuity

CFR Code of Federal Regulations
CLUE Contact Lens User Experience

COAS Complete Ophthalmic Analysis System

COM Clinical Operations Manager CRA Clinical Research Associate

CRF Case Report Form

CRO Contract Research Organization

CT Center Thickness

D Diopter

DMC Data Monitoring Committee eCRF Electronic Case Report Form EDC Electronic Data Capture

ETDRS Early Treatment Diabetic Retinopathy Study

FDA Food and Drug Administration

GCP Good Clinical Practice

HIPAA Health Insurance Portability and Accountability Act

IB Investigator's Brochure ICF Informed Consent Form

ICH International Conference on Harmonization

IDEInvestigational Device ExemptionIECIndependent Ethics CommitteeIRBInstitutional Review Board

ISO International Organization for Standardization

ITT Intent-to-Treat

JJVC Johnson & Johnson Vision Care, Inc.

LC Limbus Center

logMAR Logarithm of Minimal Angle of Resolution MedDRA<sup>©</sup> Medical Dictionary for Regulatory Activities

MOP Manual of Procedures

NIH National Institutes of Health

OD Right Eye

OHRP Office for Human Research Protections
OHSR Office for Human Subjects Research

OS Left Eye

OU Both Eyes

PD Protocol Deviation

PHI Protected Health Information

PI Principal Investigator
PIG Patient Instruction Guide
PQC Product Quality Complaint
PRO Patient Reported Outcome

QA Quality Assurance QC Quality Control

SAE Serious Adverse Event/Serious Adverse Experience

SAP Statistical Analysis Plan SAS Statistical Analysis System

SD Standard Deviation

SOP Standard Operating Procedure

UADE Unanticipated Adverse Device Effect

USADE Unanticipated Serious Adverse Device Effect

VA Visual Acuity

#### 1. INTRODUCTION AND BACKGROUND

Johnson & Johnson Vision launched their most recent multifocal contact lens called ACUVUE® OASYS MULTIFOCAL in March, 2021. The lens is recommended for presbyopes who have up to -0.75 D of refractive cylinder. There is a considerable population of presbyopic patients who have greater than -0.75 D of cylinder, in one or both eyes. Currently there are a limited number of soft toric multifocal lenses available. This study will evaluate the performance of prototype daily disposable multifocal toric lenses with a similar optical design to ACUVUE® OASYS MULTIFOCAL which are manufactured in senofilcon A (C3) material with an added high energy visible (HEV) light blocker.

#### 1.1. Name and Descriptions of Investigational Products

Test Article: JJVC Investigational Multifocal Toric Contact Lenses manufactured in Senofilcon A (C3) material with UV/HEV blocker Refer to Table 1 in Section 6.1 the protocol.

#### 1.2. Intended Use of Investigational Products

The Investigational Test lens is indicated for daily wear for the optical correction of refractive ametropia (myopia, hyperopia) and presbyopia in phakic or aphakic persons with non-diseased eyes who may need up to +2.50 D of ADD power and have astigmatism in the range of -1.00 D to -1.50 D. In this study, the lenses will be used in a population of presbyopes who require +1.25 D to +3.75 D or -1.25 D to -3.75 D of spherical correction, -1.00 D to -1.50 D of cylinder, cylinder axis within  $90^{\circ}\pm30^{\circ}$  and add powers of +0.75 D to +2.50 D (see Section 3.2).

#### 1.3. Summary of Findings from Nonclinical Studies

All previous pre-clinical findings were deemed satisfactory prior to proceeding with clinical trials on humans. For the most comprehensive nonclinical information regarding JJVC Multifocal Toric Contact Lenses manufactured in senofilcon A material refer to the latest version of the CR-6435 Investigator's Brochure.

#### 1.4. Summary of Known Risks and Benefits to Human Subjects

For the most comprehensive risk and benefit information regarding JJVC Multifocal Toric Contact Lenses manufactured in senofilcon A material refer to the latest version of the CR-6435 Investigator's Brochure and Informed Consent.

# 1.5. Relevant Literature References and Prior Clinical Data Relevant to Proposed Clinical Study

Investigational multifocal toric lenses with the same design and similar materials have been evaluated in two feasibility clinical studies prior to this study. A summary of these studies is shown below, and relevant safety information for these studies is included in the CR-6435 Investigator's Brochure.

was a single-arm dispensing evaluation of multifocal toric investigational lenses in a myopic population with against-the-rule astigmatism. Lenses used in this study had a slightly different material formulation than the lenses being used in the current CR-6435 study. The

study lenses were worn for approximately 2 weeks (with a first follow-up visit after 6-8 days, and second follow-up visit after a further 6-8 days). Forty subjects were enrolled in the study and thirty-seven completed it. No adverse events were reported.

is an ongoing single-arm dispensing evaluation of multifocal toric investigational lenses in a hyperopic population with against-the-rule astigmatism. This study is testing lenses with an older formulation (same as the one used in \_\_\_\_\_\_) in comparison with a newer formulation (same as the one to be used in the current CR-6435 study). In the 2x3 crossover study design involving 6 visits, subjects wear one of the study lens types for approximately 2 weeks, and the other study lens type for approximately 3 weeks. As of May 5, 2021, 30 subjects had been enrolled, with 3 screen failures, 2 discontinuations, 23 completed and 2 ongoing. One non-significant ocular adverse has been reported to date, which was determined to be not related to the study lens.

In addition to these two multifocal toric studies, a series of studies have been performed on a non-toric multifocal version of the study lens. Further details of the safety profile of these related lens types are included in the Investigator's Brochure.

#### 2. STUDY OBJECTIVES, ENDPOINTS AND HYPOTHESES

#### 2.1. Objectives

The main purpose of the study is to confirm the performance of the study lens relative to previously established safety and efficacy criteria. Study results may also be compared to the results obtained in other studies through aggregation of results in graphs and tables.

#### Primary Objective

The primary objective of this study is to assess the clinical performance of investigational multifocal toric contact lenses with respect to subjective vision measured via CLUE<sup>TM</sup> questionnaire, and visual acuity (logMAR) after approximately two weeks of lens wear.

#### Secondary Objective

The secondary objectives of this study are to compare the clinical performance of investigational multifocal toric contact lenses with the subjects' habitual correction with respect to subjective vision, comfort and lens handling measured via the CLUE<sup>TM</sup> questionnaire after approximately two weeks of lens wear.

#### **Exploratory Objectives**

Additional exploratory objectives are to evaluate the lens fit acceptance and toric fit of the investigational multifocal toric lenses, and the ocular health via slit lamp findings.

#### 2.2. Endpoints

Primary Endpoints
Visual Acuity (logMAR)

Multiple assessments of binocular and monocular visual acuity will be made during the study, but the binocular measurements made at the 2-week follow-up evaluation using high contrast letters in bright illuminance conditions will be the primary endpoint. At distance (4 meters), VA is assessed using ETDRS Charts; while near (40 cm) and intermediate (64 cm) assessments will be made using reduced Guillon-Poling charts. Visual acuity will be measured using high and low contrast charts in bright illuminance conditions. Visual acuity will also be measured using high contrast charts in dim illuminance conditions created by the use of goggles. See in Appendix H for details regarding the collection of visual acuity (logMAR).

#### CLUE Vision Score

Subjective quality of vision will be assessed using the Contact Lens User Experience (CLUE<sup>TM</sup>) questionnaire after approximately 2-weeks of wear. CLUE is a validated patientreported outcomes questionnaire to assess patient-experience attributes of soft, disposable contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, ages 18-65. Derived CLUE<sup>TM</sup> scores using Item Response Theory (IRT) follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response with a range of 0-120. A 5-point increase in an average CLUE<sup>TM</sup> score translates into 10% shift in the distribution of scores for population of soft contact lens wearers.<sup>5</sup>

#### Secondary Endpoints

- CLUE Vision Scores, change from baseline to 2-week follow-up
- CLUE Comfort Scores, change from baseline to 2-week follow-up
- CLUE Handling Scores, change from baseline to 2-week follow-up

#### Other Exploratory endpoints:

- Percentage of eyes with an unacceptable lens fit during the study
- Percentage of lens fits with rotation stability within 5 degrees at 15 minutes after insertion at the fitting visit
- Percentage of lens fits with absolute rotation error within 10 degrees at 15 minutes after insertion at the fitting visit
- Percentage of eyes with Grade 3 or 4 findings during the post-fit period.

#### 2.3. Hypotheses

All primary hypotheses must be met in order to satisfy the study objective.

#### Primary Hypotheses

- 1. After approximately 2 weeks of wear in the optimized lenses, the mean overall quality of vision score with the Test lens will be statistically better than 40 points on CLUE scale for myopic subjects.
- 2. After approximately 2 weeks of wear in the optimized lenses, the mean overall quality of vision score with the Test lens will be statistically better than 32 points on CLUE scale for hyperopic subjects.

- 3. After approximately 2 weeks of wear in the optimized lenses, the binocular, high-luminance, high-contrast distance (4 M) logMAR visual acuity of the test lens will be statistically better than 0.00 logMAR. This will be determined using ETDRS LogMAR acuity testing charts.
- 4. After approximately 2 weeks of wear in the optimized lenses, the binocular, high-luminance, high-contrast intermediate (64 cm) logMAR visual acuity of the test lens will be statistically better than +0.17 logMAR. This will be determined using Guillon/Poling LogMAR acuity testing charts.
- 5. After approximately 2 weeks of wear in the optimized lenses, the binocular, high-luminance, high-contrast near (40 cm) logMAR visual acuity of the test lens will be statistically better than +0.17 logMAR. This will be determined using Guillon/Poling LogMAR acuity testing charts.

Secondary Hypotheses

Secondary hypotheses will be tested for the hyperopes and the myopes separately.

- 1. After approximately 2 weeks of wear in the optimized lenses, the mean overall quality of vision CLUE score for Test lens will be non-inferior to the baseline score measured for habitual correction. A non-inferiority margin of -5 will be used.
- 2. After approximately 2 weeks of wear in the optimized lenses, the mean comfort CLUE score with the Test lens will be non-inferior to the baseline score measured for habitual correction. A non-inferiority margin of -5 will be used.
- 3. After approximately 2 weeks of wear in the optimized lenses, the mean lens handling CLUE score with the Test lens will be non-inferior to the baseline score measured for habitual correction. A non-inferiority margin of -5 will be used.

#### 3. TARGETED STUDY POPULATION

#### 3.1. General Characteristics

The population to be studied will consist of adapted contact lens wearers with presbyopia, ametropia (hyperopia or myopia) and astigmatism.

#### 3.2. Inclusion Criteria

Potential subjects must satisfy all of the following criteria to be enrolled in the study:

Inclusion Criteria following Screening The subject must:

1. Read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.

- 2. Appear able and willing to adhere to the instructions set forth in this clinical protocol.
- 3. Be at least 40 and not more than 70 years of age at the time of screening.
- 4. Own a wearable pair of spectacles if required for their distance vision.
- 5. Be an adapted soft contact lens wearer in both eyes (i.e. worn lenses for at least 8 hours per day at least two days per week for the past 4 weeks).
- 6. Be already wearing a presbyopic contact lens correction (e.g., reading spectacles over contact lenses, multifocal or monovision contact lenses, etc.) or if not respond positively to at least one symptom on the "Presbyopic Symptoms Questionnaire".

#### Inclusion Criteria at Baseline Evaluation

- 7. The subject's distance spherical component of their refraction must be in the range of either -1.25 D to -3.75 D, or +1.25 D to +3.75 D.
- 8. The subject's refractive cylinder must be -1.00 D to -1.50 D in each eye, with the cylinder axes in the range of  $90^{\circ}\pm30^{\circ}$ .
- 9. The subject's ADD power must be in the range of +0.75 D to +2.50 D in each eye.
- 10. The subject must have best corrected distance visual acuity of 20/20-3 or better in each eye.

#### 3.3. Exclusion Criteria

Potential subjects who meet any of the following criteria will be excluded from participating in the study:

Exclusion Criteria following Screening The subject must not:

- 1. Be currently pregnant or lactating.
- 2. By self-report, have any systemic disease (e.g. Sjögren's Syndrome), allergies, infectious disease (e.g., hepatitis, tuberculosis), contagious immunosuppressive diseases (e.g., HIV), autoimmune disease (e.g. rheumatoid arthritis), or other diseases, by self-report, which are known to interfere with contact lens wear and/or participation in the study.
- 3. Use systemic medications that may interfere with contact lens wear or cause blurred vision. See Section 9.1 for additional details regarding excluded systemic medications.
- 4. Currently use ocular medication (with the exception of rewetting drops).
- 5. Have any known hypersensitivity or allergic reaction to single use preservative free rewetting drops or sodium fluorescein.
- 6. Have had any previous, or have any planned, ocular or intraocular surgery (e.g. radial keratotomy, PRK, LASIK, cataract surgery, retinal surgery, etc.).
- 7. Have had previous eyelid injuries, surgeries or procedures which are known to have caused abnormal eyelid position or movement, by self-report.
- 8. Have participated in any contact lens or lens care product clinical trial within 7 days prior to study enrollment.
- 9. Be an employee or immediate family member of an employee of clinical site (e.g., Investigator, Coordinator, Technician).
- 10. Have a history of amblyopia or strabismus, by self-report.

11. Have a history of herpetic keratitis, by self-report.

Exclusion Criteria at Baseline Evaluation The subject must not:

- 12. Have ocular allergies, infections or other ocular abnormalities that are known to interfere with contact lens wear and/or participation in the study. This may include, but not be limited to entropion, ectropion, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions, aphakia, or corneal distortion
- 13. Have any Grade 3 or greater slit lamp findings (e.g., edema, corneal neovascularization, corneal staining, tarsal abnormalities, conjunctival injection) on the FDA scale.

#### 3.4. Enrollment Strategy

Study subjects will be recruited from the Institution/clinical site's subject database and/or utilizing Independent Ethics Committee (IEC) or Institutional Review Board (IRB) approved materials.

#### 4. STUDY DESIGN AND RATIONALE

#### 4.1. Description of Study Design

The study is a bilateral, single-masked, single-arm, 4-visit dispensing study. Approximately 90 (50 myopes and 40 hyperopes) subjects will be enrolled into this study with the target of completing approximately 80 (45 myopes and 35 hyperopes) subjects.

The study begins with an initial visit (Visit 1). If a subject is found to meet all eligibility criteria, the subject will be dispensed the study lens in a bilateral fashion. If the subject is dispensed study lenses at the initial visit, then three follow-up visits will occur. The first follow-up visit will occur approximately one week after the initial visit. If necessary, the lens power may be modified at Visit 2, then a new pair of lenses with the final lens power will be dispensed. The second follow-up (Visit 3) will occur approximately 1-week after Visit 2. The 3<sup>rd</sup> and final follow-up evaluation (Visit 4) will occur approximately 1-week after Visit 3.

#### 4.2. Study Design Rationale

A single-arm study was chosen to confirm the performance of the study lens relative to previously established safety and efficacy criteria. These criteria have been defined based on data from previous studies of 1-DAY ACUVUE® MOIST Multifocal (1DAMM) that have been successfully marketed since 2015.<sup>5</sup> Additionally, results from this study may be compared to data from a similar single-arm study on a marketed multifocal toric lens.<sup>7</sup> Data from these studies will be compared by creating tables and graphs of aggregate data after the study databases are all hard-locked.

#### 4.3. Enrollment Target and Study Duration

Approximately 50 myopic subjects with against-the-rule astigmatism will be enrolled, with the aim that at least 45 will complete the study. Approximately 40 hyperopic subjects with against-the-rule astigmatism will be enrolled, with the aim that at least 35 will complete the study. Subjects to be enrolled will have -1.00 D to -1.50 D of astigmatism in both eyes with  $90^{\circ}\pm30^{\circ}$  axis

Lenses in minus powers and plus powers will be evaluated in two separate phases of the study which may run at different times depending on when lenses become available. Each phase of the study will last approximately 3 months. Each individual subject is expected to be in the study for approximately 3 weeks. Lens will be worn as daily disposable and will be replaced daily.

#### 5. TEST ARTICLE ALLOCATION AND MASKING

#### 5.1. Test Article Allocation

This is a single-arm study. All subjects will be dispensed the study lens in a bilateral fashion.

#### 5.2. Masking

Subjects will be masked to the study lens to help reduce potential bias. Subjects will be unaware of the identity of the investigational product. Investigators and clinical site personnel involved in the data collection will not be masked as to the identity of the investigational product.

Under normal circumstances, the mask should not be broken until all subjects have completed the study and the database is finalized. Otherwise, the mask should be broken only if specific emergency treatment/course of action would be dictated by knowing the treatment status of the subject. In such cases, the Investigator may, in an emergency, contact the medical monitor. In the event the mask is broken, the Sponsor must be informed as soon as possible. The date, time, and reason for the unmasking must be documented in the subject record. The Investigator is also advised not to reveal the study treatment assignment to the clinical site or Sponsor personnel.

Subjects who have had their treatment assignment unmasked are expected to return for all remaining scheduled evaluations. Subjects who are discontinued may be replaced.

#### 5.3. Procedures for Maintaining and Breaking the Masking

The test articles mask shall not be broken unless information concerning the lens type is necessary for the urgent medical treatment of a subject. The Sponsor must be notified before the mask is broken.

When dispensing test articles, the following steps should be followed to maintain randomization codes:

- 1. Investigator or designee (documented on the Delegation Log) will consult the lens fitting schedule/randomization scheme to obtain the test article assignment for that subject prior to dispensing.
- 2. Investigator or designee will record the subject's number on the appropriate line of the randomization scheme
- 3. Investigator or designee will pull the appropriate test articles from the study supply. All test articles that are opened, whether dispensed (placed/fit on eye or dispensed outside the clinical site) or not, must be recorded on the Test Article Accountability Log in the "Dispensed" section.

#### 6. STUDY INTERVENTION

#### 6.1. Identity of Test Articles

The following contact lenses will be used in this study:

Table 1: Test Articles

| | Test Lens |
|--------------------------------------|---------------------------------------|
| Name | JJVC Investigational Multifocal Toric |
| | Contact Lenses manufactured in |
| | Senofilcon A (C3) material with |
| | UV/HEV blocker |
| Manufacturer | JJVC |
| Lens Material | senofilcon A(C3) with chromophore |
| Nominal Base Curve | 8.5 |
| Nominal Diameter | 14.3 |
| Nominal Distance Powers (D) | -1.00 to -4.00 in 0.25D steps, |
| | +1.00 to +4.00 in 0.25D steps |
| Nominal Cylinder Powers (D) | -1.00 |
| Cylinder axes (°) | 70, 90, 110 |
| Nominal ADD Power (D) | Low, Mid, High |
| Water Content | 38% |
| Oxygen Permeability (Dk) | 122.0 |
| Wear Schedule in Current Study | Daily Disposable |
| Replacement Frequency | Daily |
| Packaging Form (vial, blister, etc.) | Blister |

Each subject will wear approximately 42 lenses for the average 21 day dispensing period, plus any additional lenses needed for modifications and replacements.

#### 6.2. Ancillary Supplies/Products

The following solutions will be used in this study:

Table 2: Ancillary Supplies

| | Single-Use Preservative-Free Rewetting Solutions (any of these three options may be supplied) | | |
|---|---|---|---|
| Solution<br>Name/Description | Eye-Cept <sup>®</sup> Rewetting Drops | ScleralFil® Preservative Free Saline Solution | LacriPure<br>Saline Solution |
| Manufacturer | Optics<br>Laboratory | Bausch +<br>Lomb | Menicon |
| Preservative | Non-<br>Preserved | Non-<br>Preserved | Non-Preserved |

Stopwatches will be provided to research sites to help with managing the timing of toric fit assessments and lens settling.

#### 6.3. Administration of Test Articles

Test articles will be dispensed to subjects meeting all eligibility requirements, including any dispensing requirements set forth in this clinical protocol. Subjects will be dispensed an adequate supply of test articles to complete the study. Test articles which are lost or damaged may be replaced at the discretion of the Investigator.

#### 6.4. Packaging and Labeling

The test articles will be packaged in blisters as the primary packaging with an investigational lens label. The test articles will be in plastic bags as the secondary packaging form. The sample study label is shown below:



#### 6.5. Storage Conditions

Test articles will be maintained at ambient temperatures at the clinical site. Test articles must be kept under secure conditions.

#### 6.6. Collection and Storage of Samples

When possible, any lens or test article associated with an Adverse Event and/or a Product Quality Complaint must be retained and stored in a glass vial with moderate solution pending directions from the sponsor for potential return to JJVC.

#### 6.7. Accountability of Test Articles

JJVC will provide the Investigator with sufficient quantities of study articles and supplies to complete the investigation. The Investigator is asked to retain all lens shipment documentation for the test article accountability records.

Test articles must be kept in a locked storage cabinet, accessible only to those assigned by the Investigator for dispensing. The Investigator may delegate this activity to authorized study site personnel listed on the Site Delegation Log. All test articles must be accounted. This includes:

- 1. What was dispensed for the subject for trial fitting, to wear out of the office, or issued for the subject to replace appropriately between visits.
- 2. What was returned to the Investigator unused, including expired or malfunctioning product.
- 3. The number and reason for unplanned replacements.

The Investigator will collect all unused test articles from the subjects at the end of the subject's participation. Subject returned unused test articles must be separated from the clinical study inventory of un-dispensed test articles and must be labeled with the subject number and date of return. Following final reconciliation of test articles by the monitor, the Investigator or monitor will return all unused test articles to JJVC.

If there is a discrepancy between the shipment documents and the contents, contact the study monitor <u>immediately.</u>

## 7. STUDY EVALUATIONS

## 7.1. Time and Event Schedule

Table 3: Time and Events

| Visit Information | Visit 1<br>Screening, | Visit 2<br>Treatment 1 | Visit 3<br>Treatment 1 | Visit 4<br>Treatment 1 |
|---|---|---|---|---|
| | Baseline,<br>Treatment 1 | Follow-up 1 | Follow-up 2 | Follow-up 3 |
| Time Point | Day 0 | 7 ± 1 days after<br>Visit 1 | 7 ± 1 days after<br>Visit 2 | 7 ± 1 days after<br>Visit 3 |
| Estimated Visit Duration | 2.5 hours | 1.0 hours | 1.0 hours | 1.5 hours |
| Statement of Informed Consent | X | | | |
| Demographics | X | | | |
| Medical History/Concomitant<br>Medications/Review | X | | | |
| AE/Concomitant Med Review | | X | X | X |
| Habitual Contact Lens<br>Information & Wear Schedule | X | | | |
| Contact Lens History | X | | | |
| Habitual Lens Wear Time Study Lens Wear Time | X | X | X | X |
| Compliance | | X | X | X |
| Presbyopic Symptoms Ouestionnaire | X | Α | A | A |
| Screening Inclusion/Exclusion Criteria | X | | | |
| Patient Reported Outcomes | X | X | X | X |
| Ocular Symptoms | X | X | X | X |
| Subjective Acceptance | | X | X | X |
| Entrance distance and near Visual Acuity | X | X | X | X |
| Lens Removal | X | X | X | X |
| Keratometry | X | | | |
| Subjective Sphero-Cylindrical Refraction | X | | | |
| Near ADD Determination | X | | | |
| Ocular Dominance ADD Refinement | X<br>X | | | |
| Near Visual Acuity | X | | | |
| Slit Lamp Biomicroscopy | X | X | X | |
| Baseline Inclusion/ Exclusion | X | - 11 | - 11 | |
| Lens Selection | XOO | 0.0 | | |
| Right Lens Insertion | XOO | 0.0 | | |
| Right Lens 1 Minute and 3<br>Minute Rotation | XOO | 00 | | |
| Left Lens Insertion | XOO | 0.0 | | |
| Left Lens 1 Minute and 3<br>Minute Rotation | XOO | 00 | | |
| Lens Settling | XOO | 0.0 | | |
| Toric Fit Assessment | XOO | XOO | X | X |

| Visit Information | Visit 1 | Visit 2 | Visit 3 | Visit 4 |
|---|---|---|---|---|
| | Screening, | Treatment 1 | Treatment 1 | Treatment 1 |
| | Baseline, | Follow-up 1 | Follow-up 2 | Follow-up 3 |
| | Treatment 1 | | • | |
| Time Point | Day 0 | $7 \pm 1$ days after | $7 \pm 1$ days after | $7 \pm 1$ days after |
| | | Visit 1 | Visit 2 | Visit 3 |
| Estimated Visit Duration | 2.5 hours | 1.0 hours | 1.0 hours | 1.5 hours |
| Subjective Lens Fit | XOO | XOO | X | X |
| Assessment | X 0 0 | XOO | Λ | Λ |
| Visual Satisfaction | XOO | 0 0 | | |
| Study Lens Distance and Near | X O O | 0.0 | | |
| Visual Acuity | AOO | 00 | | |
| Over Refraction and Visual | XOO | XOO | X | X |
| Acuity | AOO | AOO | Λ | Λ |
| Lens Power Modification (if | X | X | | |
| required) | 71 | 71 | | |
| Additional Lens Power | | X | | |
| Modification (if required) | | 71 | | |
| Collect unworn lenses (if | | 0 | | |
| required) | | | | |
| Visual Performance | | | X | X |
| Insert new pair of lenses | | X | X | |
| Exit Snellen Distance and | X | X | X | |
| Near Visual Acuity | Λ | Λ | Λ | |
| Dispensing Criteria | X | X | X | |
| Dispensing | | X | X | |
| Subject Instructions | X | X | X | |
| Schedule Follow-Up | X | X | X | |
| Final Evaluation | | | | X |

Note: O denotes Optional items performed if required based on results

## 7.2. Detailed Study Procedures

#### VISIT 1

Subjects must report to the visit wearing their habitual contact lenses to accurately assess baseline PRO (CLUE and MRD) performance. If the subject is not wearing their lenses they must be rescheduled.

| | Visit 1: Screening | |
|---|---|---|
| Step | Procedure | Details |
| 1.1 | Statement of<br>Informed Consent | Each subject must read, understand, and sign the Statement of Informed Consent before being enrolled into the study. The Principal Investigator or his/her designee conducting the informed consent discussion must also sign the consent form. |
| | | Note: The subject must be provided a signed copy of this document. |

| Visit 1: Screening | | |
|---|---|---|
| Procedure | Details | |
| Demographics | Record the subject's year of birth, age, gender, race and ethnicity. | |
| Medical History and<br>Concomitant<br>Medications | Questions regarding the subject's medical history and concomitant medications. | |
| Habitual Contact<br>Lens Information | Questions regarding the subject's habitual lens type and parameters. | |
| Habitual Contact<br>Lens Wear Schedule | Record the duration of wearing this contact lens type and power (number of years and months). During the past four weeks, what is the minimum number of days per week that the subject has worn their lenses for at least 8 hours. | |
| Contact Lens History | Record the subject's correction type (i.e. monovision, multifocal, sphere with readers, etc.). | |
| Wear time and<br>Comfortable Wear<br>time with Habitual<br>lenses | Record the subject's wear time and comfortable wear time with their habitual contact lenses. | |
| Presbyopic<br>Symptoms<br>Questionnaire | Subjects will be asked if they are wearing a presbyopic correction and whether they are experiencing any of five common symptoms of presbyopia. | Appendix<br>E |
| Eligibility after<br>Screening | All responses to Screening Inclusion Criteria questions must be answered "yes" and all responses to Exclusion Criteria must be answered "no" for the subject to be considered eligible. If subject is deemed to be ineligible after screening, proceed to Final Evaluation and complete Subject Disposition, Refraction and | |
| | Demographics Medical History and Concomitant Medications Habitual Contact Lens Information Habitual Contact Lens Wear Schedule Contact Lens History Wear time and Comfortable Wear time with Habitual lenses Presbyopic Symptoms Questionnaire Eligibility after | Demographics Record the subject's year of birth, age, gender, race and ethnicity. Medical History and Concomitant Medications Habitual Contact Lens Information Habitual Contact Lens Wear Schedule Habitual Contact Lens Wear Schedule Record the subject's medical history and concomitant medications. Record the duration of wearing this contact lens type and parameters. Record the duration of wearing this contact lens type and power (number of years and months). During the past four weeks, what is the minimum number of days per week that the subject has worn their lenses for at least 8 hours. Contact Lens History Record the subject's correction type (i.e. monovision, multifocal, sphere with readers, etc.). Record the subject's wear time and comfortable wear time with Habitual lenses Presbyopic Symptoms Questions regarding the subject's habitual lens type and parameters. Record the duration of wearing this contact lens type and power (number of years and months). During the past four weeks, what is the minimum number of days per week that the subject has worn their lenses for at least 8 hours. Record the subject's correction type (i.e. monovision, multifocal, sphere with readers, etc.). Record the subject's wear time and comfortable wear time with their habitual contact lenses. Subjects will be asked if they are wearing a presbyopic correction and whether they are experiencing any of five common symptoms of presbyopia. All responses to Screening Inclusion Criteria questions must be answered "yes" and all responses to Exclusion Criteria must be answered "no" for the subject to be considered eligible. If subject is deemed to be ineligible after |

| | Visit 1: Baseline | |
|---|---|---|
| Step | Procedure | Details |
| 1.10 | Baseline PRO | The subject will evaluate the vision |
| | (CLUE and MRD) | characteristics, comfort characteristics, |
| | and CLDEQ-8 | handling characteristics, and visual symptoms |
| | Questionnaires | |

| | | Visit 1: Baseline | |
|---|---|---|---|
| Step | Procedure | Details Details | |
| Всер | Trocedure | of their habitual lenses using the PRO (CLUE and MRD) and CLDEQ-8 questions. | |
| 1.11 | Ocular Symptoms | Subjects will respond to a verbal open-ended symptoms questionnaire. | |
| 1.12 | Entrance Distance<br>and Near Visual<br>Acuity | Record the distance and near Snellen visual acuity (OD, OS, OU) to the nearest letter with the subject's habitual contact lenses in place. For near measurements use the ETDRS 2000 Series Chart 1 or 2. If the subject habitually wears reading glasses over their contact lenses, these may be worn for near acuity. | |
| 1.13 | Lens Removal | Have the subject remove their habitual lenses and store in an approved storage solution. | |
| 1.14 | Keratometry / SimK | Keratometry/SimK will be performed OD and OS and the steep and flat dioptric power and corresponding meridians recorded. | |
| 1.15 | Subjective Spherocylindrical Refraction | An optimal, binocular balanced distance sphero-cylindrical refraction will be performed. Record the refraction and distance visual acuity (OD, OS, OU) to the nearest letter. Note: Best distance visual acuity with sphero-cylindrical refraction must be at least 20/20 <sup>-3</sup> in each eye for the subject to be | |
| 1.16 | Near ADD<br>Determination | eligible in the study. The near reading addition will be determined using the binocular crossed cylinder technique (BCC) at 40 cm | |
| 1.17 | Ocular Dominance | Determine the distance ocular dominance with the best distance correction in place using a +1.00-blur test. If the results are equivocal use the sighting dominance test to determine the dominant eye used for the study. | Appendix<br>F |
| 1.18 | ADD Refinement | Place the BCC result in the trial frame and refine the near prescription with trial lenses (or flippers) under binocular conditions. | |
| 1.19 | Near Visual Acuity | Using the ETDRS 2000 Series Chart 1 or 2 near card placed at 40 cm. Record the near visual acuity (OD, OS, OU). | |

| | Visit 1: Baseline | |
|---|---|---|
| Step | Procedure | Details |
| 1.20 | Biomicroscopy | FDA Slit Lamp Classification Scale will be used to grade the findings and determine eligibility. |
| | | If any of these slit lamp findings are Grade 3 or higher, the subject will be discontinued. If discontinued a final examination must be completed. |
| | | If the clearance of the fluorescein needs to be expedited, preservative-free rewetting drops may be instilled. |
| 1.21 | Eligibility after<br>Baseline | All responses to Inclusion Criteria questions must be answered "yes" and all responses to Exclusion Criteria questions must be answered "no" for the subject to be considered eligible. |
| | | If subject is deemed to be ineligible after baseline, proceed to Final Evaluation and complete all forms. |

| | , | TT' '- 1 TD 1 T | |
|---|---|---|---|
| | , | Visit 1: Treatment 1 Lens Fitting | T |
| Step | Procedure | Details | |
| 1.22 | Lens Selection | Select the lens power and axis based on the | Appendix |
| | | refraction and fitting guide for each eye. | D |
| | | Record the test lens parameters (power and | |
| | | lot number). | |
| 1.23 | Right Lens Insertion | Subjects will insert the right lens themselves. | |
| | | If the lens is uncomfortable, inspect for | |
| | | damage and remove, reinsert or replace as | |
| | | necessary. | |
| | | Damaged lenses will be stored in a labeled | |
| | | vial with saline for shipment back to the | |
| | | Sponsor. Complete the Quality Product | |
| | | Complaint form. | |
| 1.24 | Timed Settling for | The investigator will start a stopwatch as | |
| | Right Lens | soon as the right lens is inserted. | |
| | | soon as the right tens is inserted. | |
| | | Note: All lenses in this study have toric | |
| | | orientation marks at the 6 and 12 o'clock | |

| | Visit 1: Treatment 1 Lens Fitting | |
|---|---|---|
| Step | Procedure | Details |
| | | positions. Rotation measurements are |
| | | made relative to a vertical reference line. |
| | | Record base nasal or base temporal rotation |
| | | to the nearest degree. |
| | | At one (1) minute after insertion: Record: |
| | | 1. The rotational position to the nearest |
| | | degree |
| | | At three (3) minutes after insertion: Record: |
| | | The rotational position to the nearest degree |
| 1.25 | Left Lens Insertion | Subjects will insert the left lens themselves. If |
| | | the lens is uncomfortable, inspect for damage |
| | | and remove, reinsert or replace as necessary. |
| | | Damaga 4 1 - 1 |
| | | Damaged lenses will be stored in a labeled |
| | | vial with saline for shipment back to the |
| | | Sponsor. Complete the Quality Product Complaint form. |
| 1.26 | Timed Settling for | The investigator will start a stopwatch as |
| 1.20 | Left Lens | soon as the left lens is inserted. |
| | Left Leffs | soon as the left lens is inserted. |
| | | Note: All lenses in this study have toric |
| | | orientation marks at the 6 and 12 o'clock |
| | | positions. Rotation measurements are |
| | | made relative to a vertical reference line. |
| | | Record base nasal or base temporal rotation |
| | | to the nearest degree. |
| | | At one (1) minute after insertion: Record: |
| | | 1. The rotational position to the nearest |
| | | degree |
| | | At three (3) minutes after insertion: Record: |
| 1.07 | T C 41 | The rotational position to the nearest degree |
| 1.27 | Lens Settling | Allow the study lenses to settle for a |
| 1.28 | Toric Fit Evaluation | minimum of 15 minutes. Record: |
| 1.28 | TOTIC TILEVALUATION | |
| | | • The rotational position to the nearest |
| | | degree |
| | | • Lens stability with blink |
| | | • Toric fit acceptable or unacceptable |
| | | Toric lens fit will be unacceptable if lenses |
| | | rotated more than 30 degrees, or lens |
| | | stability is worse than 5 degrees movement |

| | Visit 1: Treatment 1 Lens Fitting | |
|---|---|---|
| Step | Procedure | Details |
| Бієр | Troccadic | with blink. If toric fit is unacceptable, remove, store, and label the lenses, and proceed to Final Evaluation. |
| 1.29 | Lens Fit Assessment | <ul> <li>Evaluate and grade lens centration, primary gaze movement, upgaze movement and tightness (push-up test).</li> <li>The subject should not proceed to wear the lenses if any of the following is observed:</li> <li>presence of limbal exposure (appearance of clear cornea) in any gaze</li> <li>presence of edge lift</li> <li>presence of unacceptable movement (excessive or insufficient) in all three movement categories (primary gaze, upgaze, and push-up).</li> <li>If either lens is deemed unacceptable, the subject will be discontinued from the study. Remove the lenses, perform a slit-lamp evaluation, and complete the Final Evaluation form.</li> </ul> |
| 1.30 | Determine Visual<br>Satisfaction | Determine if the subject's vision is acceptable with the lenses. Allow the subject to look down a hallway or out of a window for distance vision assessments, and for them to read a book, magazine or similar for near vision. |
| 1.31 | Study Lens Distance<br>and Near Visual<br>Acuity | Record the distance and near Snellen visual acuity (OD, OS, OU) to the nearest letter with the study contact lenses in place. For near measurements use the ETDRS 2000 Series Chart 1 or 2. |
| 1.32 | Distance Over-<br>Refraction and<br>Distance Visual<br>Acuity | Perform a distance over-refraction OD and OS using loose lenses outside of the phoropter under ambient room illumination. The distance over-refraction may also be refined under binocular conditions. Record the results. The results of the distance over-refraction may also be checked for the impact on near vision under monocular and/or binocular conditions. |

| | Visit 1: Treatment 1 Lens Fitting | | |
|---|---|---|---|
| Step | Procedure | Details | |
| 1.33 | Lens Power Modification (if applicable) | If the subject reports unsatisfactory vision, or is unable to obtain 20/30 distance visual acuity OU with the lenses than a modification must be attempted. If the subject reports satisfactory vision with the lenses a modification is not required however may be made at the Investigators discretion based | Appendix<br>D |
| | | upon their findings on the measured visual acuity and/or over- refraction. Note: switching to a non-multifocal lens per Step 3 of the Fitting Guide is not an available option in this study. | |
| | | Select the reason(s) for lens change (select all that apply): • The settled lens rotation is such that one of the other available lens cylinder axis would be better (use LARS rule to determine the replacement lens cylinder axis) • Power Modification needed • Unsatisfactory Vision • Other (specify reason) | |
| | | If one or both lenses are modified, repeat steps <b>1.22 through 1.32</b> for one or both eyes as appropriate. A maximum of <i>two</i> lens modifications are allowed. | |
| 1.34 | Exit Distance and<br>Near Visual Acuity | Record the distance and near Snellen visual acuity (OD, OS, OU) to the nearest letter with the study contact lenses in place. For near measurements use the ETDRS 2000 Series Chart 1 or 2. | |
| 1.35 | Dispensing<br>Criteria | <ul> <li>The lenses may be dispensed for 6-8 days, if the following criteria are met:</li> <li>Distance Snellen acuity equal to or better than 20/30 OU</li> <li>Subject must indicate that the vision is acceptable.</li> <li>Subject must indicate that the comfort of the lenses is acceptable.</li> <li>Lenses must have an acceptable toric and general lens fit.</li> </ul> | |

| Visit 1: Treatment 1 Lens Fitting | | |
|---|---|---|
| Step | Procedure | Details |
| 1.36 | Dispensing | Only enough lenses will be dispensed to the subject to wear for the required number of days until their follow-up visit. No additional lenses will be dispensed. |
| 1.37 | Subject Instructions | Instruct the Subject on the following: The lenses will be worn on a daily disposable wear basis. Instruct the subject to bring back all unworn study lenses. Instruct the subject no cleaning or disinfecting solutions will be used for this lens type. If determined necessary by the Investigator sterile non-preserved rewetting drops may be dispensed to be used as needed for dryness. Subjects will be instructed to wear lenses for a minimum of 6 hours a day, every day between visits. One missed day of lens wear between visits is acceptable. Subjects will be instructed to wear study lenses to the next visit. It is not required that they have worn lenses for 6 hours on the day of the visit. Subjects will be instructed to wear their glasses when not wearing the study lenses. A patient instruction booklet will be provided. Note: In the event a lens is lost or damaged, the subject may return to the investigator site for a replacement. As much as reasonably possible, a damaged lens should be returned to the investigational site and then returned to the Sponsor. If lens damage is present, complete the Product Quality Complaint |
| | | Form. The lens will be stored in a labeled |
| | | vial with saline solution and returned to the Sponsor. |
| 1.38 | Schedule | The subject will be scheduled to return for |
| 1.50 | Follow-up | their follow-up appointment in 7±1 days. |
VISIT 2

The subjects must present to Visit 2 wearing the study lenses.

| | Visit 2: Treatment 1 Follow-Up 1 | |
|---|---|---|
| Step | Procedure | Details |
| 2.1 | Adverse Events and | Review any changes to the subject's medical |
| | Concomitant | history or concomitant medications from the |
| | Medications Review | previous study visit. Record any changes, |
| | | and any adverse events. |
| 2.2 | Wear time and | Record the average wearing time and |
| | Comfortable Wear | comfortable wearing time with the study |
| | time (Study Lenses) | lenses. |
| 2.3 | Compliance | Confirm compliance with the prescribed |
| | | wear schedule. |
| 2.4 | PRO (CLUE and | The subject will respond to the Follow-Up |
| 2.5 | MRD) Questionnaires | PRO (CLUE and MRD) Questionnaires. |
| 2.5 | Subject Reported | Subjects will respond to a verbal open-ended |
| 2.6 | Ocular Symptoms | symptoms questionnaire. |
| 2.6 | Subjective Acceptance | Record whether the subject's distance and |
| 2.7 | Entrance Distance and | near vision with the lenses is acceptable. Record the distance and near Snellen visual |
| 2.7 | Near Visual Acuity | acuity (OD, OS, OU) to the nearest letter with |
| | Incal visual Acuity | the study contact lenses in place. |
| | | For near measurements use the ETDRS |
| | | 2000 Series Chart 1 or 2. |
| 2.8 | Distance Over- | Perform a distance over-refraction OD and |
| 2.8 | Refraction and | OS using loose lenses outside of the |
| | Distance Visual Acuity | phoropter under ambient room illumination. |
| | Distance Visual Meanty | The distance over-refraction may also be |
| | | refined under binocular conditions. |
| | | Record the results. The results of the |
| | | distance over-refraction may also be checked |
| | | for the impact on near vision under |
| | | monocular and/or binocular conditions. |
| 2.9 | Toric Fit Evaluation | Record: |
| | | The rotational position to the nearest |
| | | degree |
| | | Lens stability with blink |
| | | Toric fit acceptable or unacceptable |
| | | Toric lens fit will be unacceptable if lenses |
| | | rotated more than 30 degrees, or lens |
| | | stability is worse than 5 degrees movement |
| | | with blink. If toric fit is unacceptable, |

| | Vi | sit 2: Treatment 1 Follow-Up 1 |
|---|---|---|
| Step | Procedure | Details |
| | | remove, store, and label the lenses, and |
| | | proceed to final evaluation. |
| 2.10 | Lens Fit Assessment | Evaluate and grade lens centration, primary |
| | | gaze movement, upgaze movement and |
| | | tightness (push-up test). |
| | | The subject should not proceed to wear the |
| | | lenses if any of the following is observed: |
| | | • presence of limbal exposure (appearance |
| | | of clear cornea) in any gaze |
| | | • presence of edge lift |
| | | • presence of unacceptable movement (excessive or insufficient) in all three |
| | | movement categories (primary gaze, |
| | | upgaze, and push-up). |
| | | 10 1 |
| | | If either lens is deemed unacceptable, the |
| | | subject will be discontinued from the study. |
| | | Remove the lenses, perform a slit-lamp |
| | | evaluation, and complete the Final Evaluation form. |
| 2.11 | Lens Power | If the subject's vision is unacceptable for at |
| 2.11 | Modification (if | least one distance or the Investigator |
| | required) | determines that the visual acuity or over- |
| | | refraction are not acceptable then a lens |
| | | modification must be made. <i>If modifications</i> |
| | | are not needed, proceed to step 2.23. |
| | | Up to <i>two</i> attempts at changes are permitted |
| | | if necessary, in order to achieve an |
| | | acceptable distance and near binocular |
| | | performance for the subject. |
| | | Select the reason(s) for lens change (select |
| | | <ul><li>all that apply):</li><li>The settled lens rotation is such that one of</li></ul> |
| | | the other available lens cylinder axis would |
| | | be better (use LARS rule to determine the |
| | | replacement lens cylinder axis) |
| | | Power Modification needed |
| | | Unsatisfactory Vision |
| | | Other (specify reason) |

| | Visit 2: Treatment 1 Follow-Up 1 | | |
|---|---|---|---|
| Step | Procedure | Details | |
| 2.12 | | Follow the fitting guide allowing for at least 10 minutes of settling time between lens changes. Note: switching to a non-multifocal lens per Step 3 of the Fitting Guide is not an available option in this study. | 11 |
| 2.12 | Lens Selection (if required) | Select the lens power, based on the Fitting Guide for each eye needing optimization. | Appendix<br>D |
| | required) | Record the test lens parameters (power and | D |
| | | lot number). | |
| 2.13 | Lens Insertion (if required) | Subjects will insert the lens themselves. If the lens is uncomfortable, inspect for damage and remove, reinsert or replace as necessary. | |
| | | Damaged lenses will be stored in labeled vial with saline solution, and clearly differentiated from the other worn lenses that will be shipped back to the Sponsor. Complete the Quality Product Complaint form. | |
| 2.14 | Timed Settling for<br>Lens (if required) | The investigator will start a stopwatch as soon as the lens is inserted. | |
| | | Note: All lenses in this study have toric orientation marks at the 6 and 12 o'clock position. Rotation measurements are made relative to a vertical reference line. Record base nasal or base temporal rotation to the nearest degree. At one (1) minute after insertion: Record: a. The rotational position to the nearest degree | |
| | | At three (3) minutes after insertion: Record: a. The rotational position to the nearest degree | |
| 2.15 | Lens Settling (if required) | Allow the study lenses to settle for a minimum of 15 minutes. | |
| 2.16 | Toric Fit Evaluation (if | Record: | |
| 2.10 | required) | • The rotational position to the nearest | |
| | | degree | |
| | | Lens stability with blink | |
| | | Lens stability with eye versions | |

| | Visit 2: Treatment 1 Follow-Up 1 | |
|---|---|---|
| Step | Procedure | Details |
| | | Toric fit acceptable or unacceptable |
| | | Toric lens fit will be unacceptable if lenses |
| | | rotated more than 30 degrees, or lens |
| | | stability is worse than 5 degrees movement |
| | | with blink. If toric fit is unacceptable, |
| | | remove, store, and label the lenses, and |
| | | proceed to final evaluation. |
| 2.17 | Lens Fit Assessment (if | Evaluate and grade lens centration, primary |
| | required) | gaze movement, upgaze movement and |
| | , | tightness (push-up test). |
| | | The subject should not proceed to wear the |
| | | The subject should not proceed to wear the lenses if any of the following is observed: |
| | | , and the second |
| | | • presence of limbal exposure (appearance of clear cornea) in any gaze |
| | | <ul> <li>presence of edge lift</li> </ul> |
| | | <ul> <li>presence of eage int</li> <li>presence of unacceptable movement</li> </ul> |
| | | (excessive or insufficient) in all three |
| | | movement categories (primary gaze, |
| | | upgaze, and push-up). |
| | | If either lens is deemed unacceptable, the |
| | | subject will be discontinued from the study. |
| | | Remove the lenses, perform a slit-lamp |
| | | evaluation, and complete the Final |
| | | Evaluation form. |
| 2.18 | Determine Visual | Determine if the subject's vision is |
| | Satisfaction (if | acceptable with the lenses. Allow the subject |
| | required) | to look down a hallway or out of a window |
| | | for distance vision assessments, and for them |
| | | to read a book, magazine or similar for near vision. |
| 2.19 | Study Lens Distance | Record the distance and near Snellen visual |
| 2.17 | and Near Visual | acuity (OD, OS, OU) to the nearest letter with |
| | Acuity (if required) | the study contact lenses in place. |
| | | For near measurements use the ETDRS 2000 |
| | | Series Chart 1 or 2. |
| 2.20 | Distance Over- | Perform a distance over-refraction OD and |
| | Refraction and | OS using loose lenses outside of the |
| | Distance Visual Acuity | phoropter under ambient room illumination. |
| | (if required) | The distance over-refraction may also be refined under binocular conditions. |
| | | remied under omocular conditions. |

| | Visit 2: Treatment 1 Follow-Up 1 | | |
|---|---|---|---|
| Step | Procedure | Details | |
| | | Record the results. The results of the | |
| | | distance over-refraction may also be checked | |
| | | for the impact on near vision under | |
| | | monocular and/or binocular conditions. | |
| 2.21 | Additional Lens Power Optimization (if required) | If the subject reports unsatisfactory vision, or is unable to obtain 20/30 distance visual acuity OU with the lenses than a modification must be attempted. If the subject reports satisfactory vision with the lenses a modification is not required however may at the Investigators discretion based upon their findings on the measured visual acuity and/or over- refraction. <i>Note:</i> switching to a non-multifocal lens per Step 3 of the Fitting Guide is not an available option in this study. | Appendix<br>D |
| | | Select the reason(s) for lens change (select all that apply): • The settled lens rotation is such that one of the other available lens cylinder axis would be better (use LARS rule to determine the replacement lens cylinder axis) • Power Modification needed • Unsatisfactory Vision • Other (specify reason) If one or both lenses are modified, repeat | |
| | | steps <b>2.13 through 2.21</b> for one or both eyes as appropriate. | |
| 2.22 | Collect unworn study lenses (if applicable) | If the lens power for either eye has been modified at this visit, collect any unworn lenses for that eye. If the subject is being discontinued for any reason, collect any unworn lenses. | |
| 2.23 | Lens Removal | Have the subject remove the study lenses. Temporarily store the worn lenses until Biomicroscopy has been completed. If no adverse event or PQC was recorded, the worn lenses may be discarded. | |
| 2.24 | Biomicroscopy | FDA Slit Lamp Classification Scale will be used to grade the findings and determine eligibility. | |

| | Visit 2: Treatment 1 Follow-Up 1 | |
|---|---|---|
| Step | Procedure | Details |
| | | If the clearance of the fluorescein needs to be expedited, preservative-free rewetting drops or saline may be instilled. |
| 2.25 | Insertion of Study<br>Lenses | Provide the subject with a <b>NEW PAIR</b> of lenses that match the power of the lenses that were removed in step 2.23 above. |
| 2.26 | Exit Distance and<br>Near Visual Acuity | Record the distance and near Snellen visual acuity (OD, OS, OU) to the nearest letter with the study contact lenses in place. For near measurements use the ETDRS 2000 Series Chart 1 or 2. |
| 2.27 | Dispensing<br>Criteria | <ul> <li>The lenses may be dispensed for 6-8 days, if the following criteria are met:</li> <li>Distance Snellen acuity equal to or better than 20/30 OU</li> <li>Subject must indicate that the vision is acceptable.</li> <li>Subject must indicate that the comfort of the lenses is acceptable.</li> <li>Lenses must have an acceptable toric and general lens fit.</li> </ul> |
| 2.28 | Dispensing | Only enough lenses will be dispensed to the subject to wear for the required number of days until their follow-up visit. No additional lenses will be dispensed. |
| 2.29 | Subject Instructions | <ul> <li>Instruct the Subject on the following:</li> <li>The lenses will be worn on a daily disposable wear basis.</li> <li>Instruct the subject to bring back all unworn study lenses.</li> <li>Instruct the subject no cleaning or disinfecting solutions will be used for this lens type.</li> <li>If determined necessary by the Investigator sterile non-preserved rewetting drops may be dispensed to be used as needed for dryness.</li> <li>Subjects will be instructed to wear lenses for a minimum of 6 hours a day, every day between visits. One missed day of lens wear between visits is acceptable.</li> </ul> |

| | Visit 2: Treatment 1 Follow-Up 1 | |
|---|---|---|
| Step | Procedure | Details |
| | | <ul> <li>Subjects will be instructed to wear study lenses to the next visit. It is not required that they have worn lenses for 6 hours on the day of the visit.</li> <li>Subjects will be instructed to wear their glasses when not wearing the study lenses.</li> </ul> |
| 2.30 | Schedule | The subject will be scheduled to return for |
| | Follow-up | their follow-up appointment in 7±1 days. |

VISIT 3

The subjects must present to Visit 3 wearing the study lenses.

| | Visit 3: Treatment 1 Follow-Up 2 | | |
|---|---|---|---|
| Step | Procedure | Details | |
| 3.1. | Adverse Events and<br>Concomitant<br>Medications Review | Review any changes to the subject's medical history or concomitant medications from the previous study visit. Record any changes, and any adverse events. | |
| 3.2. | Wear time and<br>Comfortable Wear<br>time (Study Lenses) | Record the average wearing time and comfortable wearing time with the study lenses. | |
| 3.3. | Compliance | Confirm compliance with the prescribed wear schedule. | |
| 3.4. | PRO (CLUE and MRD) and CLDEQ-8 Questionnaires | The subject will respond to the Follow-Up PRO (CLUE and MRD) and Dry Eye Questionnaires. | |
| 3.5. | Subject Reported<br>Ocular Symptoms | Subjects will respond to a verbal open-ended symptoms questionnaire. | |
| 3.6. | Subjective<br>Acceptance | Record whether the subject's distance and near vision with the lenses is acceptable. | |
| 3.7. | Entrance Distance<br>and Near Visual<br>Acuity | Record the distance and near Snellen visual acuity (OD, OS, OU) to the nearest letter with the study contact lenses in place. For near measurements use the ETDRS 2000 Series Chart 1 or 2. | |
| 3.8. | Binocular Distance<br>Over-refraction and<br>Distance Visual<br>Acuity | Perform a binocular over-refraction and record the OD and OS results and distance visual acuity. Note: No lens changes are allowed based on the over-refraction. | Appendix<br>G |

| | V | Visit 3: Treatment 1 Follow-Up 2 |
|---|---|---|
| Step | Procedure | Details |
| 3.9. | Toric Fit Evaluation | Record: |
| | | The rotational position to the nearest |
| | | degree |
| | | Lens stability with blink |
| | | _ |
| | | • Toric fit acceptable or unacceptable |
| | | Toric lens fit will be unacceptable if lenses |
| | | rotated more than 30 degrees, or lens |
| | | stability is worse than 5 degrees movement |
| | | with blink. If toric fit is unacceptable, |
| | | remove, store, and label the lenses, and |
| | | proceed to final evaluation. |
| 3.10. | Lens Fit Assessment | Evaluate and grade lens centration, primary |
| | | gaze movement, upgaze movement and |
| | | tightness (push-up test). |
| | | The subject should not proceed to wear |
| | | the lenses if any of the following is |
| | | observed: |
| | | <ul> <li>presence of limbal exposure (appearance</li> </ul> |
| | | of clear cornea) in any gaze |
| | | presence of edge lift |
| | | presence of unacceptable movement |
| | | (excessive or insufficient) in all three |
| | | movement categories (primary gaze, |
| | | upgaze, and push-up). |
| | | If either lens is deemed unacceptable, the |
| | | subject will be discontinued from the study. Remove the lenses, perform a slit-lamp |
| | | evaluation, and complete the Final |
| | | Evaluation, and complete the 1 mai |
| 3.11. | Visual Performance | Visual performance will be recorded OD, OS, |
| | Distance (4 M) | and OU for the following: |
| | Intermediate (64 cm) | Distance, Bright Illuminance |
| | Near (40 cm) | ETDRS Charts 4 M-HC#1, HC#2, HC#3 and |
| | | LC#1, LC#2 and LC#3 |
| | | Near, Bright Illuminance |
| | | Reduced Guillon-Poling Charts High Contrast |
| | | and Low Contrast Intermediate (64 cm) and |
| | | Near (40 cm). |

| | Visit 3: Treatment 1 Follow-Up 2 | |
|---|---|---|
| Step | Procedure | Details |
| | | Distance, Dim Illuminance (with <u>Distance</u> |
| | | goggles) |
| | | ETDRS Charts 4 M-HC#4, HC#5, HC#6 |
| | | Near, Dim Illuminance (with <u>Near goggles</u> ) |
| | | Reduced Guillon-Poling charts |
| | | High Contrast |
| | | Intermediate (64 cm) and Near (40 cm). |
| | | Note: |
| | | • The room illuminance must be between |
| | | 7.3 and 7.9 EV. |
| | | Distance, HC-1 Chart luminance Acceptable FV Pages 10.5.10.7. |
| | | Acceptable EV Range 10.5-10.7. • Guillon-Poling, Near Chart Luminance |
| | | Acceptable EV Range 10.8-11.1. |
| | | Do not use the Mesopic filter for Dim |
| | | luminance (Dim luminance will be |
| | | simulated by using the goggles). |
| 3.12. | Lens Removal | Have the subject remove the study lenses. |
| | | Temporarily store the worn lenses until |
| | | Biomicroscopy has been completed. If no |
| | | adverse event or PQC was recorded, the worn |
| 3.13. | Diamiaragaany | lenses may be discarded. |
| 3.13. | Biomicroscopy | FDA Slit Lamp Classification Scale will be used to grade the findings and determine |
| | | eligibility. |
| | | engionity. |
| | | If the clearance of the fluorescein needs to be |
| | | expedited, preservative-free rewetting drops |
| | | or saline may be instilled. |
| 3.14. | Insertion of Study | Provide the subject with a <b>NEW PAIR</b> of |
| | Lenses | lenses that match the power of the lenses that |
| 3.15. | Exit Distance and | were discarded in step 3.12 above. Record the distance and near Snellen visual |
| 3.13. | Near Visual Acuity | acuity (OD, OS, OU) to the nearest letter with |
| | 1 Tour Vibuar Mounty | the study contact lenses in place. |
| | | For near measurements use the ETDRS |
| | | 2000 Series Chart 1 or 2. |
| 3.16. | Dispensing | The lenses may be dispensed for 6-8 days, if |
| | Criteria | the following criteria are met: |
| | | Distance Snellen acuity equal to or better |
| | | than 20/30 OU |

| | Visit 3: Treatment 1 Follow-Up 2 | |
|---|---|---|
| Step | Procedure | Details |
| | | <ul> <li>Subject must indicate that the vision is acceptable.</li> <li>Subject must indicate that the comfort of the lenses is acceptable.</li> <li>Lenses must have an acceptable toric and general lens fit.</li> </ul> |
| 3.17. | Dispensing | Only enough lenses will be dispensed to the subject to wear for the required number of days until their follow-up visit. No additional lenses will be dispensed. |
| 3.18. | Subject Instructions | <ul> <li>Instruct the Subject on the following:</li> <li>The lenses will be worn on a daily disposable wear basis.</li> <li>Instruct the subject to bring back all unworn study lenses.</li> <li>Instruct the subject no cleaning or disinfecting solutions will be used for this lens type.</li> <li>If determined necessary by the Investigator sterile non-preserved rewetting drops may be dispensed to be used as needed for dryness.</li> <li>Subjects will be instructed to wear lenses for a minimum of 6 hours a day, every day between visits. One missed day of lens wear between visits is acceptable.</li> <li>Subjects will be instructed to wear study lenses to the next visit. It is not required that they have worn lenses for 6 hours on the day of the visit.</li> <li>Subjects will be instructed to wear their glasses when not wearing the study lenses.</li> <li>Subjects will be instructed to bring their spectacles with distance vision correction, or their habitual contact lenses to the final visit.</li> </ul> |
| 3.19. | Schedule | The subject will be scheduled to return for |
| | Follow-up | their follow-up appointment in 7±1 days. |

VISIT 4

The subjects must present to Visit 4 wearing the study lenses.

| | Visit 4: Treatment 1 Follow-Up 3 | | |
|---|---|---|---|
| Step | Procedure | Details | |
| 4.1. | Adverse Events and<br>Concomitant<br>Medications Review | Review any changes to the subject's medical history or concomitant medications from the previous study visit. Record any changes, and any adverse events. | |
| 4.2. | Wear time and<br>Comfortable Wear<br>time (Study Lenses) | Record the average wearing time and comfortable wearing time with the study lenses. | |
| 4.3. | Compliance | Confirm compliance with the prescribed wear schedule. | |
| 4.4. | Collect unworn lenses (if applicable) | The subject will return any unworn lenses. | |
| 4.5. | PRO (CLUE and MRD) and CLDEQ-8 Questionnaires | The subject will respond to the Follow-Up PRO (CLUE and MRD) and Dry Eye Questionnaires. | |
| 4.6. | Subject Reported<br>Ocular Symptoms | Subjects will respond to a verbal open-ended symptoms questionnaire. | |
| 4.7. | Subjective<br>Acceptance | Record whether the subject's distance and near vision with the lenses is acceptable. | |
| 4.8. | Entrance Distance<br>and Near Visual<br>Acuity | Record the distance and near Snellen visual acuity (OD, OS, OU) to the nearest letter with the study contact lenses in place. For near measurements use the ETDRS 2000 Series Chart 1 or 2. | |
| 4.9. | Binocular Distance<br>Over-refraction and<br>Distance Visual<br>Acuity | Perform a binocular over-refraction and record the OD and OS results and distance visual acuity. Note: No lens changes are allowed based on the over-refraction. | Appendix<br>G |
| 4.10. | Toric Fit Evaluation | <ul> <li>Record:</li> <li>The rotational position to the nearest degree</li> <li>Lens stability with blink</li> <li>Toric fit acceptable or unacceptable Toric lens fit will be unacceptable if lenses rotated more than 30 degrees, or lens stability is worse than 5 degrees movement with blink. If toric fit is unacceptable, remove, store, and label the lenses, and</li> </ul> | |

| | Visit 4: Treatment 1 Follow-Up 3 | |
|---|---|---|
| Step | Procedure | Details |
| | | proceed to final evaluation. |
| 4.11. | Lens Fit Assessment | Evaluate and grade lens centration, primary gaze movement, upgaze movement and tightness (push-up test). • The subject should not proceed to wear the lenses if any of the following is |
| | | <ul> <li>observed:</li> <li>presence of limbal exposure (appearance of clear cornea) in any gaze</li> <li>presence of edge lift</li> <li>presence of unacceptable movement (excessive or insufficient) in all three movement categories (primary gaze, upgaze, and push-up).</li> </ul> |
| | | If either lens is deemed unacceptable, the subject will be discontinued from the study. Remove the lenses, perform a slit-lamp evaluation, and complete the Final Evaluation form. |
| 4.12. | Visual Performance<br>Distance (4M)<br>Intermediate (64 cm)<br>Near (40 cm) | Visual performance will be recorded OD, OS, and OU for the following: Distance, Bright Illuminance ETDRS Charts 4M-HC#1, HC#2, HC#3 and LC#1, LC#2 and LC#3 Near, Bright Illuminance Reduced Guillon-Poling Charts High Contrast and Low Contrast Intermediate (64 cm) and Near (40 cm). |
| | | Distance, Dim Illuminance (with <u>Distance</u> goggles) ETDRS Charts 4M-HC#4, HC#5, HC#6 Near, Dim Illuminance (with <u>Near</u> goggles) Reduced Guillon-Poling charts High Contrast Intermediate (64 cm) and Near (40 cm). Note: The room illuminance must be between 7.3 and 7.9 EV. |

| | Visit 4: Treatment 1 Follow-Up 3 | |
|---|---|---|
| Step | Procedure | Details |
| | | <ul> <li>Distance, HC-1 Chart luminance Acceptable EV Range 10.5-10.7.</li> <li>Guillon-Poling, Near Chart Luminance Acceptable EV Range 10.8-11.1.</li> <li>Do not use the Mesopic filter for Dim luminance (Dim luminance will be simulated by using the goggles).</li> </ul> |
| 4.13. | Lens Removal | Have the subject remove the study lenses. Temporarily store the worn lenses until Biomicroscopy has been completed. If no adverse event or PQC was recorded, the worn lenses may be discarded. |

#### FINAL EVALUATION

The final evaluation will ordinarily take place immediately following the last scheduled follow-up visit per the study protocol. It may also take place at any point the subject discontinues the study or is terminated from the study.

| | Final Evaluation | |
|---|---|---|
| Step | Procedure | Details |
| F.1 | Final Exam Form | Indicate if the subject completed the study successfully. If subject discontinued from the study, indicate the reason. |
| F.2 | Biomicroscopy | FDA Slit Lamp Classification Scale will be used to grade the findings and determine eligibility. If the clearance of the fluorescein needs to be expedited, preservative-free rewetting drops or saline may be instilled. |
| F.3 | Subjective<br>spherocylindrical<br>Refraction | An optimal, binocular balanced distance sphero-cylindrical refraction will be performed. Record the refraction and distance visual acuity (OD, OS, OU) to the nearest letter. |
| F.4 | Exit Distance Visual Acuity | Record the distance Snellen visual acuity (OD, OS, OU) to the nearest letter, and the type of visual correction being worn (habitual lenses, distance spectacles or unaided). |

#### 7.3. Unscheduled Visits

If, during the investigation, a subject requires an unscheduled visit to the clinical site, the following information will be collected at a minimum:

- Chief complaint prompting the visit. If the reason is an adverse event, the applicable eCRF for the adverse event must be completed and subject record completed as appropriate
- Date and time of the visit and all procedures completed at the unscheduled visit
- Review of adverse event and concomitant medications
- Documentation of any test article dispensed or collected from the subject, if applicable
- Slit lamp findings (using the Slit Lamp Classification Scale)

If the Investigator withdraws a subject from the study, the final study visit case report forms must be completed indicating the reason(s) why the subject was withdrawn. The subject record must be completed documenting the date and primary reason for withdrawal and the study CRA notified.

Any ocular and non-ocular Adverse Events that are ongoing at the time of the study visit will be followed by the Investigator, within licensure, until they have resolved, returned to pretreatment status, stabilized, or been satisfactorily explained. If further treatment i.e., beyond licensure is required, the subject will be referred to the appropriate health care provider.

The following information will be collected during an unscheduled visit.

| | Unscheduled Visit | |
|---|---|---|
| Step | Procedure | Details |
| U.1 | Reason for | Indicate if the only reason for the visit is that |
| | unscheduled visit | the subject requires additional test articles. If |
| | | the reason is other than resupply of |
| | | previously dispensed lenses, specify the |
| | | reason for the visit. |
| U.2 | Chief Complaints (if | Record the subject's chief complaints for |
| | applicable) | reasons for the unscheduled visit. |
| U.3 | Adverse Events and | Review any changes to the subject's medical |
| | Concomitant | history or concomitant medications from the |
| | Medications Review | previous study visit. Record any changes, and |
| | (if applicable) | any adverse events. |
| U.4 | Entrance VA (if | Record the distance Snellen visual acuity |
| | applicable) | (OD, OS, OU) to the nearest letter, and the |
| | | type of visual correction being worn (study |
| | | lenses, habitual lenses, distance spectacles or |
| | | unaided). |
| U.5 | Subjective Sphero- | Perform bare-eye subjective spherocylindrical |
| | cylindrical | refraction with a phoropter (adopt the |
| | Refraction (if | maximum plus to maximum visual acuity |
| | applicable) | (MPMVA) approach and use the duo-chrome |

| _ | Unscheduled Visit | |
|---|---|---|
| Step | Procedure | Details |
| Бюр | Troccure | test for binocular balancing) and record the best corrected distance visual acuity to the nearest letter (OD, OS). |
| U.6 | Slit Lamp<br>Biomicroscopy (if<br>applicable) | FDA Slit Lamp Classification Scale will be used to grade the findings. If the clearance of the fluorescein needs to be expedited, preservative-free rewetting drops may be instilled. |
| U.7 | Dispensing (if applicable) | If the subject requires additional lenses to complete the wear period and is eligible to do so, provide additional lenses per the dispensing instructions given in the detailed study procedures. |
| U.8 | Toric Fit Evaluation (if applicable) | <ul> <li>After lens settling, record:</li> <li>The rotational position to the nearest degree</li> <li>Lens stability with blink</li> <li>Lens stability with eye versions</li> <li>Toric fit acceptable or unacceptable</li> <li>Toric lens fit will be unacceptable if lenses rotated more than 30 degrees, or lens stability is worse than 5 degrees movement with blink. If toric fit is unacceptable, remove, store, and label the lenses, and proceed to final evaluation.</li> </ul> |
| U.9 | Lens Fit Assessment (if applicable) | Evaluate and grade lens centration, primary gaze movement, upgaze movement and tightness (push-up test). • The subject should not proceed to wear the lenses if any of the following is observed: • presence of limbal exposure (appearance of clear cornea) in any gaze • presence of edge lift • presence of unacceptable movement (excessive or insufficient) in all three movement categories (primary gaze, upgaze, and push-up). If either lens is deemed unacceptable, the subject will be discontinued from the study. |

| | Unscheduled Visit | |
|---|---|---|
| Step | Procedure | Details |
| | | Remove the lenses, perform a slit-lamp |
| | evaluation, and complete the Final | |
| | | Evaluation form. |
| U.10 | Exit Visual Acuity | Record the distance Snellen visual acuity |
| | (if applicable) | (OD, OS, OU) to the nearest letter, and the |
| type of visual correction being | | type of visual correction being worn (study |
| | | lenses, habitual lenses, distance spectacles or |
| | | unaided). |

#### 7.4. Laboratory Procedures

None

#### 8. SUBJECTS COMPLETION/WITHDRAWAL

#### 8.1. Completion Criteria

Subjects are considered to have completed the study if they:

- provided informed consent.
- are eligible.
- completed all visits

#### 8.2. Withdrawal/Discontinuation from the Study

A subject will be withdrawn from the study for any of the following reasons:

- Subject death during the study period.
- Subject withdrawal of consent.
- Subject not compliant to protocol
- Subject lost to follow-up.
- Subject no longer meets eligibility criteria (e.g. the subject becomes pregnant).
- Subject develops significant or serious adverse events causing discontinuation of study lens wear.
- Subjects who have experienced a Corneal Infiltrative Event (CIE).
- Investigator's clinical judgment regarding the subject safety reasons (that it is in the best interest of the subject to stop treatment).
- Subject missed any study visit.
- Subject not compliant with study lens wear schedule.
- Subject not successfully dispensed due to lack of efficacy and safety including poor vision, poor comfort or unacceptable fit.

For discontinued subjects, the Investigator will:

- Complete the current visit (scheduled or unscheduled).
- Complete the Final Evaluation, indicating the reason that the subject was discontinued from the study.
- Record the spherocylindrical refraction with best corrected distance visual acuity.
- Collect used test article(s) (worn or brought to the visit) from the subject and discard them, unless otherwise stated in Section 7.2.
- Collect all unused test article(s) from the subject.
- Make arrangements for subject care, if needed, due to their study participation

An additional subject may be enrolled if a subject discontinues from the study prematurely.

In cases where a subject is lost to follow-up, every possible effort must be made to contact the subject and determine the reason for discontinuation/withdrawal. The measures taken to follow up must be documented including two written attempts and a certified letter (or equivalent) as the final attempt.

#### 9. PRE-STUDY AND CONCOMITANT INTERVENTION/MEDICATION

Concomitant medications will be documented during screening and updated during the study. Disallowed medications and therapies are medications or therapies that contraindicate contact lens wear. See the Exclusion criteria for specific details.

#### 9.1. Systemic Medications

Certain systemic medications are known to have a higher likelihood to interfere with contact lens wear, chiefly by disrupting the tear film. A summary of disallowed medications is shown in Table 4. Subjects with a history of taking these medications will be allowed to enroll only if:

• The medications have been taken on a continual or routine basis for at least 6 months and the subject has demonstrated successful contact lens wear during this time.

Or

• The subject previously used these medications on a temporary basis and has ceased that medication at least 1 week prior to signing the informed consent.

Table 4: Disallowed systemic medications

| Class of Drug | Common Indication(s) | Common Examples |
|---|---|---|
| Anticholinergics | Irritable bowel syndrome, Parkinson's disease, peptic ulcer, cystitis, nasal congestion, cold symptoms, overactive bladder, COPD | Bentyl, Spiriva, Atrovent,<br>Hyosyne, Levsin, Symax<br>Fastab, Symax SL, Homax SL,<br>Cogentin, Transderm Scop, etc. |
| Oral Phenothiazines | Antipsychotic disorders (schizophrenia, mania) | Compazine, Mellaril,<br>Thorazine, Phenergan, etc. |

| Class of Drug | Common Indication(s) | Common Examples |
|---|---|---|
| Oral/Inhaled<br>Corticosteroids | Arthritis, colitis, asthma,<br>bronchitis, allergic or<br>inflammatory conditions | Cortisone, Prednisone, Hydrocortisone, Medrol, Kenalog, Flonase etc. |
| Oral Retinoids | Seborrhea, acne | Isotretinoin, Acitretin,<br>Alitretinoin, etc. |
| Oral Tetracycline | Urinary Tract Infection, acne, chlamydia, gonorrhea | Sumycin, Achromycin V, etc. |

#### 10. DEVIATIONS FROM THE PROTOCOL

Investigator will notify study sponsor upon identification of a protocol deviation. Protocol deviations must be reported to the sponsor within 24 hours after discovery of the protocol deviation. The Investigator will report deviations per IRB/IEC requirements. All deviations will be tracked, and corrective actions implemented as appropriate.

If it becomes necessary for the Investigator to implement a deviation in order to eliminate an immediate hazard to the trial subject, the Investigator may implement the deviation immediately without notification to the sponsor. Within 24 hours after the implemented deviation, the Investigator must notify and provide the rationale to the Sponsor and, as required, the IEC/IRB.

If the deviation potentially impacts the safety of patient or changes the technical integrity of the study, then it must be reported to IEC/IRB. This is a "Major Deviation". Deviations that contradict the information contained in the Informed Consent/Assent forms will be considered Major Deviations.

Minor deviations have no substantive effect on patient safety or technical integrity of the study. They are often logistical in nature.

Protocol waivers are prohibited.

Table 5 lists examples of deviations that will constitute major and minor protocol deviations for this study.

Table 5: Examples of major and minor protocol deviations

| <b>Deviation category</b> | Major deviation | Minor deviation |
|---|---|---|
| Out-of-window visit | Visit attended 3 or more days out of visit window defined in study procedures | Visit attended 2 or fewer days out of visit window defined in study procedures |
| Insufficient wear of study lenses | Subject does not wear study lenses for at least 6 hours per day for 3 or more days between scheduled visits. | Subject does not wear study lenses for at least 6 hours per day for 2 days between scheduled visits. |

#### 11. STUDY TERMINATION

If more than 2 subjects in the investigational soft contact lens group develop serious expected (e.g., definite or probable MK) or unexpected device related adverse events, the study will be suspended. Upon review and consultation with IRB, DMC, and JJVC Safety Review committee, the study may be terminated. This potential stopping rule is established based on our trial involving approximately 200 subjects wearing the investigational soft contact lens for up to 3 years with an assumed MK rate that is below 0.2% per patient-year. The rate of 0.2% per patient year is the established rate for extended wear lenses in adults, which was requested by the FDA as a criterion for evaluating a contact lens for pediatric use in an FDA response to a pre-IDE submission. To be conservative, 200 independent patient years were used in the calculation. The probability of observing 2 cases or more incidents of MK is 0.061, and 3 cases or more incidents of MK is 0.007 (given an MK rate of 0.2% per patient year).

The occurrence of one or more Unanticipated Serious Adverse Device Effect (USADE), or any SAE where the relationship to study agent cannot be ruled out, may result in stopping further dispensing of test article. In the event of a USADE or SAE, the Sponsor may unmask the treatment regimen for the subject(s) and will discuss this with the Investigator before any further subjects are enrolled.

The Sponsor will determine when a study will be stopped. The Principal Investigator always has the discretion to initiate stopping the study based on patient safety or if information indicates the study's results are compromised.

JJVC reserves the right to terminate the study at any time for any reason. Additionally, the IEC/IRB reserves the right to terminate the study if an unreasonable risk is determined. The study can be terminated by the Principal Investigator at the individual clinical site due to specific clinical observations, if in their opinion, after a discussion with JJVC, it is determined that it would be unwise to continue at the clinical site.

JJVC (and the IEC/IRB and DMC, if applicable) will evaluate all adverse events. If it is determined that an adverse event presents an unreasonable risk, the investigation, or that part of the investigation presenting the risk, will be terminated as soon as possible.

Should the study be terminated (either prematurely or as scheduled), the Investigator will notify the IEC/IRB and Regulatory Authority as required by local regulatory requirements.

#### 12. PROCEDURE FOR HANDLING PRODUCT QUALITY COMPLAINTS

A Product Quality Complaint (PQC) refers to any written, electronic, or oral communication that alleges deficiencies related to the identity, quality, durability, reliability, safety, effectiveness or performance of test articles after they have been released for clinical trial use.

Potential complaints may come from a variety of sources including but not limited to subjects, clinical research associates (CRA), clinical operations managers (COM), medical monitors, and site personnel, etc. The following are not considered product quality complaints:

- Subject satisfaction inquiries reported via "Subjective Questionnaires" and "Patient Reported Outcomes (PRO)."
- Clinical test articles that are stored improperly or damaged after receipt at the investigational site.
- Lens replacements that occur due to drops/fall-outs.
- Damage deemed by clinicians or clinical staff to be caused by handling by the user, and not indicative of a quality deficiency (i.e. tears, rips, etc.), only in situations where there is no deficiency alleged by the subject.

Within 24 hours of site personnel becoming aware that a PQC has occurred, the PQC must be recorded in the EDC system, which will trigger an automatic email notification to the appropriate COM/CRA and Clinical QA representative. In cases where the EDC system in use is not configured to send automatic notifications or when an EDC system is not used, the COM/CRA is responsible for notifying Clinical QA upon discovery that a PQC has occurred.

Upon receipt of the EDC notification, the COM/CRA will contact the study site to collect additional information which will include:

- Date the complaint was received/recorded in the EDC System (Date of Sponsor Awareness).
- Who received the complaint.
- Study number.
- Clinical site information (contact name, site ID, telephone number).
- Lot number(s).
- Unique Subject Identifier(s).
- Indication of who first observed complaint (site personnel or subject).
- OD/OS indication, along with whether the lens was inserted.
- Any related AE number if applicable.
- Detailed complaint description (scheduled/unscheduled visit, wear time, symptoms, resolution of symptoms, etc.).
- Eve Care Provider objective (slit lamp) findings if applicable.

• Confirmation of product availability for return (and tracking information, if available), or rationale if product is not available for return

Once a complaint is received, it will be assessed by the COM, CRA, or trained site personnel to determine if it is an Adverse Event/Serious Adverse Event (AE/SAE). If the complaint results in an AE/SAE, the COM/CRA, or trained site personnel will follow Section 13 of this protocol. If the AE/SAE was potentially the result of a product quality related deficiency, these procedures also applies and will be executed in parallel.

In some cases, a PQC form may be generated in EDC by the site in error. In this event, the PQC forms will be marked "Intentionally Left Blank" or "ILB". Justification for ILB must be documented.

#### 13. ADVERSE EVENTS

#### 13.1. Definitions and Classifications

**Adverse Event (AE)** – An AE is "any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users or other persons, whether or not related to the investigational medical device."

**Note**: This definition includes events related to the investigational medical device or the comparator, and to the procedures involved. For users or other persons, this definition is restricted to events related to investigational medical devices.<sup>1</sup>

An AE includes any condition (including a pre-existing condition) that:

- 1. Was not present prior to the study, but appeared or reappeared following initiation of the study.
- 2. Was present prior to the study but worsened during the study. This would include any condition resulting from concomitant illnesses, reactions to concomitant medications, or progression of disease states.

**Note**: Pregnancy must be documented as an adverse event and must be reported to the clinical monitor and to the Sponsor immediately upon learning of the event.

Serious Adverse Event (SAE) – An SAE is any adverse event that led to any of the following:

- Death
- Serious deterioration in the health of the subject that resulted in any of the following:
- Life-threatening illness or injury
- Permanent or persistent impairment of a body structure or a body function
- Hospitalization or prolongation of patient hospitalization
- Medical or surgical intervention to prevent life-threatening illness or injury or permanent impairment to a body structure or a body function.
- Chronic disease
- Foetal distress, foetal death or a congenital physical or mental impairment of birth defect.

Diagnoses and conditions that are considered Ocular Serious Adverse Events include, but not limited to:

- Microbial Keratitis (MK)
- Iritis (including cells in the anterior chamber)
- Permanent decrease in best spectacle corrected visual acuity equivalent to 2 acuity lines or greater
- Central Corneal Opacity
- Central Corneal Neovascularization
- Uveitis
- Endophthalmitis
- Hypopyon
- Hyphemia
- Penetration of Bowman's Membrane
- Persistent Epithelial Defect
- Limbal cell Damage leading to Conjunctivalization

**Significant Adverse Events** – are defined as events that are symptomatic and warrant discontinuation (temporary or permanent) of the contact lens wear

Diagnoses and conditions that are considered Ocular Significant Adverse Events include, but not limited to the following:

- Contact Lens Induced Peripheral Ulcer (CLPU)
- Significant Infiltrative Events (SIE)
- Superior Epithelial Arcuate Lesions (SEALs)
- Any Temporary Loss of > 2 Lines of BSCVA
- Other grade 3 or higher corneal findings, such as abrasions or edema
- Non-contact lens related corneal events e.g. Epidemic Keratoconjunctivitis (EKC)
- Asymptomatic Corneal Scar
- Any corneal event which necessitates temporary lens discontinuation > 2 weeks

**Non-Significant Adverse Events** – are defined as those events that are usually asymptomatic and usually do not warrant discontinuation of contact lens wear but may cause a reduction in wear time. However, the Investigator may choose to prescribe treatment as a precautionary measure.

Diagnoses and conditions that are considered Ocular Non-Significant Adverse Events include, but not limited to the following:

- Non-significant Infiltrative Event (NSIE)
- Contact Lens Papillary Conjunctivitis (CLPC)
- Superficial Punctate Keratitis (SPK)
- Conjunctivitis: Bacterial, Viral, Allergic
- Blepharitis
- Meibomianitis
- Contact Dermatitis

- Localized Allergic Reactions
- Any corneal event not explicitly defined as serious or significant adverse event, which necessitates temporary lens discontinuation < 2 weeks

**Adverse Device Effect (ADE)** – An ADE is an "adverse event related to the use of an investigational medical device."

**Note 1**: This definition includes adverse events resulting from insufficient or inadequate instructions for use, deployment, implantation, installation, or operation, or any malfunction of the investigational medical device.

**Note 2**: This definition includes any event resulting from use error or from intentional misuse of the investigational medical device.<sup>1</sup>

**Unanticipated Adverse Device Effect (UADE)** – A UADE is any serious adverse effect on health or safety or any life-threatening problem or death caused by, or associated with, the test article, if that effect, problem, or death was not previously identified in nature, severity, or degree of incidence in the investigational plan, Investigator's Brochure or protocol, or any other unanticipated serious problem associated with the test article that relates to the rights, safety and welfare of subjects.

#### 13.2. Assessing Adverse Events

In conjunction with the medical monitor, the Investigator will evaluate adverse events to ensure the events are categorized correctly. Elements of categorization will include:

- Seriousness/Classifications (see definition in section 13.1).
- Causality or Relatedness i.e. the relationship between the test article, study treatment or study procedures and the adverse event (not related, unlikely related, possibly related, or related see definition in Section 13.2.1).
- Adverse Event Severity Adverse event severity is used to assess the degree of intensity of the adverse event (mild, moderate, or severe see definition in Section 13.2.2).
- Outcome not recovered or not resolved, recovering or resolving, recovered or resolved with sequelae, recovered or resolved, death related to adverse event, or unknown.
- Actions Taken none, temporarily discontinued, permanently discontinued, or other.

#### 13.2.1. Causality Assessment

**Causality Assessment** – A determination of the relationship between an adverse event and the test article. The test article relationship for each adverse event should be determined by the investigator using these explanations:

- Not Related- An adverse event that is not related to the use of the test article, study treatment or study procedures.
- Unlikely Related An adverse event for which an alternative explanation is more likely, e.g. concomitant treatment, concomitant disease(s), or the relationship of time suggests that a causal relationship is not likely.

- Possibly Related An adverse event that might be due to the use of the test article, or to the study treatment or study procedures. An alternative explanation, e.g. concomitant treatment, concomitant disease(s), is inconclusive. The relationship in time is reasonable. Therefore, the causal relationship cannot be excluded.
- Related An adverse event that is listed as a possible adverse effect (device) or adverse reaction (drug) and cannot be reasonably explained by an alternative explanation, e.g. concomitant treatment of concomitant disease(s). The relationship in time is very suggestive, e.g. it is confirmed by de-challenge and re-challenge.

#### 13.2.2. Severity Assessment

**Severity Assessment** – A qualitative assessment of the degree of intensity of an adverse event as determined by the Investigator or reported to him/her by the subject. The assessment of severity is made irrespective of test article, study treatment or study procedure relationship or seriousness of the event and should be evaluated according to the following scale:

- Mild Event is noticeable to the subject but is easily tolerated and does not interfere with the subject's daily activities.
- Moderate Event is bothersome, possible requiring additional therapy, and may interfere with the subject's daily activities.
- Severe Event is intolerable, necessitates additional therapy or alteration of therapy and interferes with the subject's daily activities.

#### 13.3. Documentation and Follow-Up of Adverse Events

The recording and documenting of adverse events (ocular and non-ocular) begin when the subjects are exposed to the test article, study treatment or study procedure. Adverse events reported before the use of test article, start of study treatment, or study procedures will be recorded as medical history. However, if the condition deteriorates at any time during the study it will be recorded and reported as an AE. Untoward medical events reported after the subject's exit from the study will be recorded as adverse events at the discretion of the Investigator.

Upon finding an adverse event, the Principal Investigator will document the condition in the subject record and in the eCRFs and complete the Adverse Event eCRF.

Complete descriptions of all adverse events must be available in the subject record. All Adverse Events including local and systemic reactions not meeting the criteria for "serious adverse events" shall be captured on the appropriate case report form or electronic data system. All adverse events occurring while the subject is enrolled in the study must be documented appropriately regardless of relationship.

It is the Investigator's responsibility to maintain documentation of each reported adverse event. All adverse events will be followed in accordance with applicable licensing requirements. Such documentation will include the following:

- Adverse event (diagnosis not symptom).
- Drawings or photographs (where appropriate) that detail the finding (e.g., size, location, and depth, etc.).

- Date the clinical site was notified.
- Date and time of onset.
- Date and time of resolution.
- Adverse event classification, severity, and relationship to test articles, as applicable.
- Treatment regimen instituted (where appropriate), including concomitant medications prescribed, in accordance with applicable licensing requirements.
- Any referral to another health care provider if needed.
- Outcome, ocular damage (if any).
- Likely etiology.
- Best corrected visual acuity at the discovery of the event and upon conclusion of the event, if the AE is related to the visual system.

Upon discovery of an AE that is deemed 'possibly related' or 'related' to the test article or study procedures (whether related to the visual system or not), an AE review form must be completed. Additional dated and initialed entries should be made at follow-up evaluations. Separate forms must be completed for each eye if the AE is bilateral.

In addition, if an infiltrate(s) is present, he/she will complete the Corneal Infiltrate Assessment eCRF. Where necessary, a culture of the corneal lesion will be collected to determine if the infection is microbial in nature. If cultures are collected, the date of culture collection and laboratory utilized will be recorded.

Changes in the severity of an AE shall be documented to allow an assessment of the duration of the event at each level of intensity to be performed. Adverse events characterized as intermittent require documentation of the onset and duration of each episode. Changes in the assessment of relationship to the Test Article shall also be clearly documented.

Subjects who present with an adverse event shall be followed by the Investigator, within licensure, until all signs and symptoms have returned to pre-treatment status, stabilized, or been satisfactorily resolved. If further treatment beyond licensure is required, the patient will be referred to the appropriate health care provider. The Investigator will use his/her clinical judgment as to whether a subject reporting with an adverse event will continue in the study. If a subject is discontinued from the study, it will be the responsibility of the Investigator to record the reason for discontinuation. The Investigator will also document the adverse event appropriately and complete the Adverse Event eCRF. Any subjects with ongoing adverse events related to the test article, study treatment or study procedures, as of the final study visit date, should be followed to resolution of the adverse event or until referral to an appropriate health care provider, as recommended by the Investigator. Non-ocular adverse events that are not related to the test article, study treatment, or study procedures may be recorded as "ongoing" without further follow-up.

#### 13.4. Reporting Adverse Events

The Investigator will notify the Sponsor of an adverse event by e-mail, facsimile, or telephone as soon as possible and no later than 24 hours from discovery for any serious /significant adverse events, and 2 days from discovery for any non-significant adverse event. In addition,

a written report will be submitted by the Principal Investigator to the IEC/IRB according to their requirements (Section 13.4.2). The report will comment whether the adverse event was considered to be related to the test article, study treatment or study procedures.

#### 13.4.1. Reporting Adverse Events to Sponsor

#### Serious/Significant Adverse Events

The Investigator will inform the sponsor of all serious/significant adverse events occurring during the study period as soon as possible by e-mail or telephone, but no later than 24 hours following discovery of the event. The Investigator is obligated to pursue and obtain information requested by the Sponsor in addition to that information reported on the eCRF. All subjects experiencing a serious/significant adverse event must be followed up and all outcomes must be reported.

When medically necessary, the Investigator may break the randomization code to determine the identity of the treatment that the subject received. The Sponsor and study monitor should be notified prior to unmasking the test articles.

In the event of a serious/significant adverse event, the Investigator must:

- Notify the Sponsor immediately.
- Obtain and maintain in the subject's records all pertinent medical information and medical judgment for colleagues who assisted in the treatment and follow-up of the subject.
- Provide the Sponsor with a complete case history which includes a statement as to whether the event was or was not related to the use of the test article.
- Notify the IEC/IRB as required by the IEC/IRB reporting procedure according to national regulations.

#### **Unanticipated (Serious) Adverse Device Effect (UADE)**

In the event of an Unanticipated (Serious) Adverse Device Effect (UADE), the Investigator will submit a report of the UADE to the Sponsor and IEC/IRB as soon as possible, but no later than 24 hours after the Investigator first learns of the effect. This report is in addition to the immediate notification mentioned above.

The Sponsor must conduct an evaluation of the UADE and must report the results of the evaluation to FDA, the IEC/IRB and participating Investigators within 10 working days after the Sponsor first receives notification of the effect.

#### **Non-Serious Adverse Events**

All non-serious adverse events, including non-serious adverse device effects, will be reported to the sponsor by the Investigator no later than 2 days from discovery.

#### 13.4.2. Reporting Adverse Events to the Responsible IEC/IRB and Health Authorities

Adverse events that meet the IEC/IRB requirements for reporting must be reported within the IEC/IRB's written guidelines. Each clinical site will refer to and follow any guidelines set forth

by their Approving IEC/IRB. Each clinical site will refer to and follow any guidelines set forth by their local governing Health Authorities.

The Sponsor will report applicable Adverse Events to the local health authorities according the written guidelines, including reporting timelines.

#### 13.5. Event of Special Interest

None

#### 13.6. Reporting of Pregnancy

Subjects reporting pregnancy (by self-report) during the study will be discontinued after the event is recorded as an Adverse Event. Once discontinued, pregnant participants and their fetuses will not be monitored for study related purposes. Pregnant participants are not discontinued from contact lens or solution related studies for safety concerns, but due to general concerns relating to pregnancy and contact lens use. Specifically, pregnant women are discontinued due to fluctuations in refractive error and/or visual acuity that occur secondary to systemic hormonal changes, and not due to unforeseen health risks to the mother or fetus.

#### 14. STATISTICAL METHODS

#### 14.1. General Considerations

Statistical Analysis will be undertaken by the sponsor or under the authority of the sponsor. A general description of the statistical methods to be implemented in this clinical trial is outlined below.

All data summaries and statistical analyses will be performed using the Statistical Analysis System (SAS) software Version 9.4 or higher (SAS Institute, Cary, NC).<sup>8</sup> Throughout the analysis of data, the results for each subject/eye will be used when available for summarization and statistical analysis. Unscheduled visits will be summarized separately and will be excluded from the statistical analysis.

Summary tables (descriptive statistics and/or frequency tables) will be provided for all baseline variables, efficacy variables and safety variables as appropriate. Continuous variables will be summarized with descriptive statistics (n, mean, standard deviation [SD], median, minimum and maximum). Frequency count and percentage of subjects or eyes within each category will be provided for categorical data.

#### 14.2. Sample Size Justification

This study was designed and powered to demonstrate that the binocular high luminance high contrast, visual performance (logMAR) of the Test lens at distance (4 meters), intermediate (64 cm) and near (40 cm) after 2-week of lens wear in the optimized lenses is superior to 0.00, +0.17 and +0.17 logMAR, respectively. Additionally, this study was also powered to show that CLUE vision scores for the Test lens for the hyperopic population is greater than 32 points and greater than 40 points for the myopic population. The sample size calculation included

two historical studies, and Previous hyperopic data was not available for the Test lens, therefore, data from was used because it evaluated lenses with a similar lens design on a hyperopic population. Data from was used for the myopic population since this study evaluated lenses with the same lens design and similar material as the current Test lens on a population of myopic subjects.

Table 6: Historical Binocular High Luminance High Contrast Visual Performance – 2-Week Follow-up

| <b>Chart Position</b> | Mean | SD* | Minimum | Maximum |
|-----------------------|--------|--------|---------|---------|
| Distance (4 M) | -0.048 | 0.0943 | -0.220 | 0.280 |
| Intermediate (64 cm) | -0.015 | 0.1183 | -0.240 | 0.320 |
| Near (40 cm) | 0.097 | 0.1318 | -0.200 | 0.500 |

<sup>\*</sup>SD: Standard Deviation

Table 7: Historical CLUE Scores – 2-Week Follow-up

| CLUE Domain | Strata | Baseline | 2-Week Follow-up |
|-------------|----------|-------------|------------------|
| | | Mean (SD*) | Mean (SD*) |
| Vision | Hyperope | 45.5(14.71) | 47.3(18.65) |
| | Myope | 42.9(15.43) | 55.1(20.73) |
| Comfort | Hyperope | 50.7(19.70) | 60.9(22.38) |
| | Myope | 54.5(20.39) | 62.7(21.95) |
| Handling | Hyperope | 50.9(17.26) | 56.6(21.12) |
| | Myope | 56.9(16.49) | 70.6(18.02) |

<sup>\*</sup>SD: Standard Deviation

Sample size calculations for each primary endpoint were carried out using a 2-sided one sample mean t-test, with a family wise error rate of 5%. The calculation was performed using the POWER<sup>11</sup> procedure in SAS Version 9.4<sup>8</sup>. The Bonferroni<sup>12</sup> method was used to adjust the type I error for multiple primary hypotheses  $\alpha = \frac{0.05}{5} = 0.01$ . A power analysis was also performed for each secondary hypothesis to test for non-inferiority of the 2-week follow-up relative to the baseline assessment with respect to CLUE vision, comfort and handling scores. The power analysis was performed for each secondary hypothesis separately using the POWER procedure and 2-sided t-test for paired means with alpha=0.05. The power Analysis was performed for different scenarios of intraclass correlation and effect sizes. The sample size required for all primary endpoints is displayed in Table 8, while the power analysis for the secondary endpoints is located in Table 9.

<sup>\*\*</sup>This summary included data from both

Table 8: Sample Size Estimates for Primary Endpoints

| Endpoint | Power | Sample Size |
|--------------------------------------|-------|-------------|
| Visual Acuity - Distance (4 M) | 80.6% | 42 |
| Visual Acuity - Intermediate (64 cm) | 80.1% | 7 |
| Visual Acuity - Near (40 cm) | 80.7% | 36 |
| CLUE Vision Scores – Hyperopes | 80.1% | 18 |
| CLUE Vision Scores – Myopes | 80.9% | 22 |

Table 9: Power Analysis for Secondary Endpoints

| Endpoint | Strata | correlation | Effect size | Power |
|-----------------|------------------|-------------|-------------|-------|
| Vision – CFB* | Hyperope<br>N=35 | 0.3 | 1 | 42.3% |
| | | | 3 | 75.0% |
| | | 0.5 | 1 | 65.5% |
| | | | 3 | 86.0% |
| | Myope<br>N=45 | 0.3 | 3 | 78.1% |
| | | | 5 | 91.7% |
| | | 0.5 | 3 | 88.2% |
| | | | 5 | 97.1% |
| Comfort – CFB* | Hyperope<br>N=35 | 0.3 | 3 | 58.4% |
| | | | 5 | 75.0% |
| | | 0.5 | 3 | 70.8% |
| | | | 5 | 86.3% |
| | Myope<br>N=45 | 0.3 | 3 | 67.8% |
| | | | 5 | 83.9% |
| | | 0.5 | 3 | 80.1% |
| | | | 5 | 92.9% |
| Handling – CFB* | Hyperope<br>N=35 | 0.3 | 3 | 64.8% |
| | | | 5 | 81.2% |
| | | 0.5 | 3 | 76.9% |
| | | | 5 | 90.8% |
| | Myope<br>N=45 | 0.3 | 3 | 82.6% |
| | | | 5 | 94.3% |
| | | 0.5 | 3 | 92.0% |
| | | | 5 | 98.5% |

<sup>\*</sup>CFB = Change from baseline (calculated as 2-week follow-up minus baseline)

Represents conservative power estimate based on the most conservative effect size and intraclass correlation.

While only 42 subjects are required to complete the study based on the sample size calculation, the plan is to compare the data from this study to another study which is similar in design and sample size and is assessing a marketed multifocal toric lens. Therefore, the sample size was increased in order to perform a meta-analysis at a later date. Moreover, as shown in Table 9, a

target completion of 80 subjects demonstrates a reasonable statistical power for the secondary endpoints under most of the assessed scenarios.

The plan is to enroll 90 eligible subjects with a target completion of 80 subjects (45 myopes and 35 hyperopes). During the enrollment period, the subject drop-out rate will be closely monitored, if an unexpectedly high dropout rate is observed, then the targeted total enrollment number maybe be increased accordingly to ensure that the target numbers of 45 myopes and 35 hyperopes subjects complete the study.

#### 14.3. Analysis Populations

#### **Safety Population:**

All subjects who were administered any test article excluding subjects who drop out prior to administering any test article. At least one observation should be recorded.

#### **Per-Protocol Population:**

All subjects who have successfully completed all visits and did not substantially deviate from the protocol as determined by the trial cohort review committee prior to database hard lock (Per-Protocol Population). Justification of excluding subjects with protocol deviations in the Per-Protocol Population set will be documented in a memo to file.

#### **Intent-to-Treat (ITT) Population:**

All randomized subjects regardless of actual treatment and subsequent withdrawal from study or deviation from protocol. At least one observation should be recorded.

#### 14.4. Level of Statistical Significance

All planned primary analyses for this study will be conducted with a 2-sided type I family wise error rate of 5%. The Bonferroni<sup>12</sup> method will be used to adjust for the number of primary hypotheses tested. Secondary hypotheses will be tested separately with a 2-sided type I error rate of 5% individually.

#### 14.5. Primary Analysis

#### **CLUE Vision Scores**

Vision scores after approximately 2-weeks in the optimized lenses will be analyzed using a linear mixed model. Baseline vision scores, event (visit 1: baseline, visit 2: 1-wk non-optimized, visit 3: 1-wk optimized and visit 4: 2-wk optimized), strata (hyperope and myope) and the interaction between event and strata will be included in the model as fixed effects. Other covariates such as age, gender and add power may be included when appropriate. Site will be included as a random effect (G-side). Residual errors between measurements within the same subject across event will be model using one of the following:

- Unstructured (UN)
- Compound Symmetric (CS)

• Heterogenous Compound Symmetric (CSH)

The structure that returns the lowest corrected Akaike's Information Criterion (Keselman et al. 1998)<sup>13</sup> will be selected as the structure that best fits the data. The Kenward and Roger method will be used for the calculation of the denominator of degrees of freedom.<sup>14</sup>

#### Primary hypothesis 1:

The null and alternative hypothesis for CLUE vision to test for superiority of the Test lens relative to the pre-defined threshold of 40 for myopes is as follows:

$$H_o$$
:  $\mu_{Test} \le 40$   
 $H_A$ :  $\mu_{Test} > 40$ 

Superiority will be declared if the lower limit of the 95% confidence interval of the adjusted mean for the Test lens is greater than 40. i.e.  $P(\mu_{Test} > 40) \ge 0.975$ .

#### Primary hypothesis 2:

The null and alternative hypothesis for CLUE vision to test for superiority of the Test lens relative to the pre-defined threshold of 32 hyperopes is as follows:

$$H_o$$
:  $\mu_{Test} \le 32$   
 $H_A$ :  $\mu_{Test} > 32$ 

Superiority will be declared if the lower limit of the 95% confidence interval of the adjusted mean for the Test lens is greater than 32. i.e.  $P(\mu_{Test} > 32) \ge 0.975$ .

#### **LogMAR Visual Acuity**

Binocular, high luminance, high contrast visual acuity on logMAR scale after approximately 2-weeks in the optimized lenses will be analyzed using a linear mixed model. Position(distance/intermediate/near) will be included as the only fixed effect. Site will be included as random effect (G-side). Other baseline characteristics known of importance such as age, gender and add power may be included as covariates when appropriate. The covariance between residual errors from the same subject across different positions will be selected based on the finite-sample corrected Akaike's Information Criterion (Keselman et al. 1998). Covariance structures considered may include: Homogenous compound symmetry (CS) and Unstructured covariance structure (UN). The structure that returns the lowest Akaike Information Criteria Corrected (AICC) will be selected as the structure that best fit the data. The Kenward and Roger method will be used for the calculation of the denominator of degrees of freedom. Acres of the calculation of the denominator of degrees of freedom.

#### Primary hypothesis 3:

The null and alternative hypothesis for binocular distance HLHC visual performance to test for superiority of the Test lens relative to the pre-defined threshold of 0 logMAR is as follows:

$$H_o$$
:  $\mu_{Test} \ge 0 \log MAR$   
 $H_A$ :  $\mu_{Test} < 0 \log MAR$ 

Superiority will be declared if the upper limit of the 95% confidence interval of the adjusted mean for the Test lens is below 0 logMAR. i.e.  $P(\mu_{Test} < 0) \ge 0.975$ .

#### Primary hypothesis 4:

The null and alternative hypothesis for binocular near HLHC visual performance to test for superiority of the Test lens relative to the pre-defined threshold of 0.17 logMAR is as follows:

$$H_o$$
:  $\mu_{Test} \ge 0.17 \log MAR$   
 $H_A$ :  $\mu_{Test} < 0.17 \log MAR$ 

Superiority will be declared if the upper limit of the 95% confidence interval of the adjusted mean for the Test lens is below 0.17 logMAR. i.e.  $P(\mu_{Test} < 0.17) \ge 0.975$ .

#### Primary hypothesis 5:

The null and alternative hypothesis for binocular distance HLHC visual performance to test for superiority of the Test lens relative to the pre-defined threshold of 0.17 logMAR is as follows:

$$H_o$$
:  $\mu_{Test} \ge 0.17 \log MAR$   
 $H_A$ :  $\mu_{Test} < 0.17 \log MAR$ 

Superiority will be declared if the upper limit of the 95% confidence interval of the adjusted mean for the Test lens is below 0.17 logMAR. i.e.  $P(\mu_{Test} < 0.17) \ge 0.975$ .

#### 14.6. Secondary Analysis

#### **CLUE Vision, Comfort and Handling Scores**

Vision, Comfort and Handling scores after approximately 2-weeks in the optimized lenses will be analyzed separately using a linear mixed model. event (visit 1: baseline, visit 2: 1-wk non-optimized, visit 3: 1-wk optimized and visit 4: 2-wk optimized), strata (hyperope and myope) and the interaction between event and strata will be included in the model as fixed effects. Other covariates such as age, gender and add power may be included when appropriate. Site will be included as a random effect (G-side). Residual errors between measurements within the same subject across event will be model using one of the following:

- Unstructured (UN)
- Compound Symmetric (CS)
- Heterogenous Compound Symmetric (CSH)
- Spatial Power (SP(POW))

The structure that returns the lowest corrected Akaike's Information Criterion (Keselman et al. 1998)<sup>13</sup> will be selected as the structure that best fits the data. The Kenward and Roger method will be used for the calculation of the denominator of degrees of freedom.<sup>14</sup>

#### **Hypothesis Testing**

The null and alternative hypotheses for non-inferiority are as follows and will be conducted separately for each strata (hyperopes and myopes) and CLUE vision, comfort and handling:

$$H_0$$
:  $\Delta \le -5$   
 $H_0$ :  $\Delta > -5$ 

Where  $\Delta$  is the change from baseline to 2-week follow-up (2-week follow up minus baseline). Non-inferiority of the 2-week follow-up CLUE score relative to the baseline CLUE scores of subjects' habitual lens was concluded if the lower limit of the 95% CI was above -5 (Pr: 2 – wk minus baseline > -5, ) > 0.975.

#### 14.7. Other Exploratory Analyses

Unacceptable lens fitting, Grade 3 + SLFs, absolute rotation and stability will be descriptively summarized by event (baseline, 1-wk follow-up non-optimized, 1-wk follow-up optimized and 2-wk follow-up optimized), when applicable. If unacceptable lens fitting, Grade 3 + SLFs, rotation stability > 5 degrees and absolution rotation > 10 degrees are observed during the study, then an analysis maybe conducted at the discretion of the study responsible clinician.

#### 14.8. Interim Analysis

Lenses in minus powers and plus powers will be evaluated in two separate phases of the study which may run at different times depending on when lenses become available. The study lenses for hyperopic subjects are likely to be available before the lenses for the myopic subjects. Therefore, a planned interim read will be performed once all hyperopic subjects have completed the study. The interim read will include descriptive summaries of all primary and secondary endpoints. Additionally, summaries for adverse events, lens fitting, lens rotation and stability will also be provided.

#### 14.9. Procedure for Handling Missing Data and Drop-Outs

Missing or spurious values will not be imputed. The count of missing values will be included in the summary tables and listings.

Subject dropout is expected to be one of the main reasons of missing data in this clinical trial.

Past clinical trials don't provide the evidence that subject dropout is systematic or not-at random. To evaluate the impact of missing data, sensitivity analysis will be conducted using multiple imputation methods if the proportion of subject dropout is greater than the 15%. The SAS/STAT procedures PROC MI and PROC MIANALYZE will be utilized with a parametric regression method used to make at least 15 imputations.

#### 14.10. Procedure for Reporting Deviations from Statistical Plan

The analysis will be conducted according to that specified in above sections. There are no known reasons for which it is planned to deviate from these analysis methods. If for any reason a change is made, the change will be documented in the study report along with a justification for the change.

#### 15. DATA HANDLING AND RECORD KEEPING/ARCHIVING

#### 15.1. Electronic Case Report Form/Data Collection

The data for this study will be captured on electronic case report forms (eCRFs) using an EDC system (Bioclinica). An authorized data originator will enter study data into the eCRFs using the EDC system. Data collected on equipment that is not captured in EDC will be formatted to the specification of the JJVC database manager and sent to JJVC for analysis.

The clinical data will be recorded on dedicated eCRFs specifically designed to match the study procedures for each visit. Only specifically delegated staff can enter data on a CRF. Once completed, the eCRFs will be reviewed for accuracy and completeness and signed by the Investigator. The sponsor or sponsor's representatives will be authorized to gain access to the subject recordation for the purposes of monitoring and auditing the study.

Edit checks, electronic queries, and audit trails are built into the system to ensure accurate and complete data collection. Data will be transmitted from the clinical site to a secure central database as forms are completed or updated, ensuring information accuracy, security, and confidentiality. After the final database lock, the Investigator will be provided with Individual Patient Profiles (IPP) including the full audit trail on electronic media in PDF format for all of the study data. The IPP must be retained in the study files as a certified copy of the source data for the study.

The content and structure of the eCRFs are compliant with ISO14155:2011.<sup>1</sup>

#### 15.2. Subject Record

At a minimum, subject record should be available for the following:

- subject identification
- eligibility
- study identification
- study discussion
- provision of and date of informed consent
- visit dates

- results of safety and efficacy parameters as required by the protocol
- a record of all adverse events
- follow-up of adverse events
- medical history and concomitant medication
- test article receipt/dispensing/return records
- date of study completion
- reason for early discontinuation of test article or withdrawal from the study, if applicable

The subject record is the eCRF or an external record. The author of an entry in the subject record must be identifiable. The first point of entry is considered to be the source record.

Adverse event notes must be reviewed and initialed by the Investigator.

#### 15.3. Trial Registration on ClinicalTrials.gov

This study will be registered on ClinicalTrials.gov based on the following: The purpose of the study is for design confirmation, not feasibility.

#### 16. DATA MANAGEMENT

#### 16.1. Access to Source Data/Document

The Investigator/Institution will permit trial-related monitoring, audits, IEC/IRB review and regulatory inspection(s) by providing direct access to source data/documents. Should the clinical site be contacted for an audit by an IEC/IRB or regulatory authority, JJVC must be contacted and notified in writing within 24 hours.

#### 16.2. Confidentiality of Information

Information concerning the investigational product and patent application processes, scientific data or other pertinent information is confidential and remains the property of JJVC. The Investigator may use this information for the purposes of the study only. It is understood by the Investigator that JJVC will use information developed in this clinical study in connection with the development of the investigational product and therefore may disclose it as required to other clinical investigators and to regulatory agencies. In order to allow the use of the information derived from this clinical study, the Investigator understands that he/she has an obligation to provide complete test results and all data developed during this study to the Sponsor.

#### 16.3. Data Quality Assurance

Steps will be taken to ensure the accuracy and reliability of data, include the selection of qualified investigators and appropriate clinical sites and review of protocol procedures with the Principal Investigator. The Principal Investigator, in turn, must ensure that all Sub-

Investigators and clinical site personnel are familiar with the protocol and all study-specific procedures and have appropriate knowledge of the study article.

Training on case report form completion will be provided to clinical site personnel before the start of the study. The Sponsor will review case report forms for accuracy and completeness remotely during the conduct of the study, during monitoring visits, and after transmission to data management. Any data discrepancies will be resolved with the Investigator or designee, as appropriate.

Quality Assurance representatives from JJVC may visit clinical sites to review data produced during the study and to access compliance with applicable regulations pertaining to the conduct of clinical trials. The clinical sites will provide direct access to study-related source data/documents and reports for the purpose of monitoring and auditing by JJVC and for inspection by local and regulatory authorities.

#### 16.4. Data Monitoring Committee (DMC)

Not applicable.

#### 17. CLINICAL MONITORING

The study monitors will maintain close contact with the Principal Investigator and the Investigator's designated clinical site personnel. The monitor's responsibilities will include:

- Ensuring that the investigation is being conducted according to the protocol, any subsequent versions, and regulatory requirements are maintained.
- Ensuring the rights and wellbeing of subjects are protected.
- Ensuring adequate resources, including facilities, laboratories, equipment, and qualified clinical site personnel.
- Ensuring that protocol deviations are documented with corrective action plans, as applicable.
- Ensuring that the clinical site has sufficient test article and supplies.
- Clarifying questions regarding the study.
- Resolving study issues or problems that may arise.
- Reviewing of study records and source documentation verification in accordance with the monitoring plan.

#### 18. ETHICAL AND REGULATORY ASPECTS

#### 18.1. Study-Specific Design Considerations

Potential subjects will be fully informed of the risks and requirements of the study and, during the study, subjects will be given any new information that may affect their decision to continue participation. Subjects will be told that their consent to participate in the study is voluntary and may be withdrawn at any time with no reason given and without penalty or loss of benefits to which they would otherwise be entitled. Only subjects who are fully able to understand the
risks, benefits, and potential adverse events of the study, and provide their consent voluntarily will be enrolled.

#### 18.2. Investigator Responsibility

The Principal Investigator is responsible for ensuring that the clinical study is performed in accordance with the signed agreement, the investigational plan, Section 4 of the ICH E6 guidelines on Good Clinical Practice (GCP),<sup>2</sup> and applicable regulatory requirements. GCP is an international ethical and scientific quality standard for designing, conducting, recording, and reporting studies that involve the participation of human subjects. Compliance with this standard provides public assurance that the rights, safety, and well-being of study subjects are protected, consistent with the principles of the Declaration of Helsinki 64<sup>th</sup> WMA General Assembly 2013<sup>3</sup> and that the clinical study data are credible. The Investigator must maintain clinical study files in accordance with Section 8 of the ICH E6 guidelines on Good Clinical Practice (GCP),<sup>2</sup> and applicable regulatory requirements.

### 18.3. Independent Ethics Committee or Institutional Review Board (IEC/IRB)

Before the start of the study, the Investigator (or Sponsor when applicable) will provide the IEC/IRB with current and complete copies of the following documents (where applicable):

- Final protocol.
- Sponsor-approved informed consent form (and any other written materials to be provided to the subjects)
- Investigator's Brochure (or equivalent information).
- Sponsor-approved subject recruitment materials.
- Information on compensation for study-related injuries or payment to subjects for participation in the study.
- Investigator's curriculum vitae, clinical licenses, or equivalent information (unless not required, as documented by IEC/IRB).
- Information regarding funding, name of the Sponsor, institutional affiliations, other potential conflicts of interest, and incentives for subjects.
- Any other documents that the IEC/IRB requests to fulfill its obligation.

This study will be undertaken only after IEC/IRB has given full approval of the final protocol, the informed consent form, applicable recruiting materials, and subject compensation programs, and the Sponsor has received a copy of this approval. This approval letter must be dated and must clearly identify the documents being approved.

During the study, the Investigator (or Sponsor when applicable) will send the following documents to the IEC/IRB for their review and approval, where appropriate:

- Protocol revisions
- Revision(s) to informed consent form and any other written materials to be provided to subjects
- If applicable, new or revised subject recruitment materials approved by the Sponsor
- Revisions to compensation for study-related injuries or payment to subjects for participation in the study

- Investigator's Brochure revisions
- Summaries of the status of the study (at least annually or at intervals stipulated in guidelines of the IEC/IRB)
- Reports of adverse events that are serious, unanticipated, and associated with the test articles, according to the IRB's requirements
- New information that may adversely affect the safety of the subjects or the conduct of the study
- Major protocol deviations as required by the IEC/IRB
- Report of deaths of subjects under the Investigator's care
- Notification if a new Investigator is responsible for the study at the clinical site
- Any other requirements of the IEC/IRB

For protocol revisions that increase subject risk, the revisions and applicable informed consent form revisions must be submitted promptly to the IEC/IRB for review and approval before implementation of the change(s).

At least once a year, the IEC/IRB will review and reapprove this clinical study. This request should be documented in writing.

At the end of the study, the Investigator (or Sponsor where required) will notify the IEC/IRB about the study completion. Documentation of this notification must be retained at the clinical site and a copy provided to the CRO or Sponsor as applicable.

#### 18.4. Informed Consent

Each subject or their representative, must give written consent according to local requirements after the nature of the study has been fully explained. The consent form must be signed before performance of any study-related activity. The consent form that is used must be approved by both the Sponsor and by the reviewing IEC/IRB. The informed consent is in accordance with principles that originated in the Declaration of Helsinki,<sup>3</sup> current ICH<sup>2</sup> and ISO 14155<sup>1</sup> guidelines, applicable regulatory requirements, and Sponsor Policy.

Before entry into the study, the Investigator or an authorized member of the clinical site personnel must explain to potential subject the aims, methods, reasonably anticipated benefits, and potential hazards of the study, and any discomfort it may entail. Subjects will be informed that their participation is voluntary and that they may withdraw consent to participate at any time.

The subject will be given sufficient time to read the informed consent form and the opportunity to ask questions. After this explanation and before entry into the study, consent should be appropriately recorded by means of the subject's dated signature. After having obtained the consent, a copy of the informed consent form must be given to the subject.

Each subject for this study will complete an assent and a parent or legal guardian must give written informed consent according to local requirements after the nature of the study has been fully explained. The assent and consent forms must be signed before performance of any study-related activity. The assent and consent forms that are used must be approved by both the

Sponsor and by the reviewing IEC/IRB. The assent and informed consent forms should be in accordance with principles that originated in the Declaration of Helsinki, 3 current ICH<sup>2</sup> and GCP guidelines, applicable regulatory requirements, and Sponsor policy. Before entry into the study or pre-screening, the Investigator or an authorized member of the clinical site personnel must explain to the potential subject and parent and/or legal guardian the aims, methods, reasonably anticipated benefits, and potential hazards of the study or pre-screening, and any discomfort it may entail. Subjects and parent and/or legal guardian will be informed that their participation is voluntary and that they may withdraw consent to participate at any time. They will be informed that choosing not to participate will not affect the care the subject will receive. Finally, they will be told that the Investigator will maintain a subject identification register for the purposes of long-term follow-up if needed and that their records may be accessed by health authorities and authorized Sponsor personnel without violating the confidentiality of the subject, to the extent permitted by the applicable law(s) or regulations. By signing the assent and informed consent form, the subject is authorizing such access and agrees to be contacted after study completion by health authorities and authorized Sponsor personnel for the purpose of obtaining consent for additional safety evaluations if needed.

### 18.5. Privacy of Personal Data

The collection, processing and disclosure of personal data and medical information related to the Study Subject, and personal data related to Principal Investigator and any clinical site personnel (e.g., name, clinic address and phone number, curriculum vitae) is subject to compliance with the Health Information Portability and Accountability Act (HIPAA) in the United States<sup>15</sup> and other applicable personal data protection and security laws and regulations. Appropriate measures will be employed to safeguard these data, to maintain the confidentiality of the person's related health and medical information, to properly inform the concerned persons about the collection and processing of their personal data, to grant them reasonable access to their personal data and to prevent access by unauthorized persons.

All information obtained during the course of the investigation will be regarded as confidential. All personal data gathered in this trial will be treated in strictest confidence by Investigators, monitors, Sponsor's personnel and IEC/IRB. No data will be disclosed to any third party without the express permission of the subject concerned, with the exception of Sponsor personnel (monitor, auditor), IEC/IRB and regulatory organizations in the context of their investigation related activities that, as part of the investigation will have access to the CRFs and subject records.

The collection and processing of personal data from subjects enrolled in this study will be limited to those data that are necessary to investigate the efficacy, safety, quality, and utility of the investigational product(s) used in this study.

These data must be collected and processed with adequate precautions to ensure confidentiality and compliance with applicable data privacy protection laws and regulations.

The Sponsor ensures that the personal data will be:

• processed fairly and lawfully.

- collected for specified, explicit, and legitimate purposes and not further processed in a way incompatible with these purposes.
- adequate, relevant, and not excessive in relation to said purposes.
- accurate and, where necessary, kept current.

Explicit consent for the processing of personal data will be obtained from the participating subject before collection of data. Such consent should also address the transfer of the data to other entities and to other countries.

The subject has the right to request through the Investigator access to his personal data and the right to request rectification of any data that are not correct or complete. Reasonable steps should be taken to respond to such a request, taking into consideration the nature of the request, the conditions of the study, and the applicable laws and regulations.

Appropriate technical and organizational measures to protect the personal data against unauthorized disclosures or access, accidental or unlawful destruction, or accidental loss or alteration must be put in place. Sponsor personnel whose responsibilities require access to personal data agree to keep the identity of study subjects confidential.

#### 19. STUDY RECORD RETENTION

In compliance with the ICH/GCP guidelines,<sup>2</sup> the Investigator/Institution will maintain all CRFs and all subject records that support the data collected from each subject, as well as all study documents as specified in ICH/GCP<sup>2</sup> and all study documents as specified by the applicable regulatory requirement(s). The Investigator/Institution will take measures to prevent accidental or premature destruction of these documents.

Essential documents must be retained until at least two (2) years after the last approval of a marketing application in an ICH region and until there are no pending or contemplated marketing applications in an ICH region or until at least two (2) years have elapsed since the formal discontinuation of clinical development of the investigational product. These documents will be retained for a longer period if required by the applicable regulatory requirements or instructed by the Sponsor. It is the responsibility of the Sponsor to inform the Investigator/Institution as to when these documents no longer need to be retained.

If the responsible Investigator retires, relocates, or for other reasons withdraws from the responsibility of keeping the study records, custody must be transferred to a person who will accept the responsibility. The Sponsor must be notified in writing of the name and address of the new custodian. Under no circumstance shall the Investigator relocate or dispose of any study documents before having obtained written approval from the Sponsor.

If it becomes necessary for the Sponsor or the appropriate regulatory authority to review any documentation relating to this study, the Investigator must permit access to such reports. If the Investigator has a question regarding retention of study records, he/she should contact JJVC.

#### 20. FINANCIAL CONSIDERATIONS

Remuneration for study services and expenses will be set forth in detail in the Clinical Research Agreement. The Research Agreement will be signed by the Principal Investigator and a JJVC management representative prior to study initiation.

JJVC reserves the right to withhold remuneration for costs associated with protocol violations such as:

- Continuing an ineligible subject in the study.
- Scheduling a study visit outside the subject's acceptable visit range.

JJVC reserves the right to withhold final remuneration until all study related activities have been completed, such as:

- Query resolution.
- Case Report Form signature.
- Completion of any follow-up action items.

#### 21. PUBLICATION

There is no plan to publish the outcome of this investigation.

#### 22. REFERENCES

- 1. ISO 14155:2011: Clinical Investigation of Medical Devices for Human Subjects Good Clinical Practice. Available at: https://www.iso.org/standard/45557.html
- 2. International Conference on Harmonization Good Clinical Practice E6 (ICH-GCP). Available at: http://www.ich.org/products/guidelines/efficacy/article/efficacy-guidelines.html
- 3. Declaration of Helsinki Ethical principles for Medical Research Involving Human Subjects. Available at: https://www.wma.net/policies-post/wma-declaration-of-helsinki-ethical-principles-for-medical-research-involving-human-subjects/
- 4. United States (US) Code of Federal Regulations (CFR). Available at: https://www.gpo.gov/fdsys/browse/collectionCfr.action?collectionCode=CFR
- 5. Wirth RJ, et al. Development of the Contact Lens User Experience: CLUE Scales. *Optom Vis Sci.* 2016;93(8):801-808
- 6. Karkkainen T. Clinical Study Report v3.0. An Evaluation of the Performance of the Vistakon Investigational Multifocal Contact Lens. 31 March, 2015.
- 7. Franklin R. Clinical Study Protocol v2.0. Evaluation of Visual Acuity with a Reusable Toric Multifocal Contact Lens. 10 February 2021.
- 8. SAS Institute Inc: SAS® 9.4 Statements: Reference TEC, NC: SAS Institute Inc; 2014.
- 9. Karkkainen T. Clinical Study Report, v2.0. Evaluation of a Novel Toric Multifocal Contact Lens in Hyperopic Presbyopes. 27 December, 2017.
- 10. Franklin R. Clinical Study Report, v1.0. Pilot Evaluation of a Silicone Hydrogel Daily Disposable Toric Multifocal Contact Lens. 15 March, 2021.
- 11. SAS Institute Inc. 2016 SAS/STAT® 14.3 User's Guide. Cary NC: SAS Institute Inc.

- 12. Bonferroni C. Calculation of the insurance groups of heads. *Studies in Honour of Professor Salvatore Ortu Carboni*. 1935;Rome: Italy:13-60.
- 13. Keselman HJ, Algina J, Kowalchuk RK, Wolfinger RD. A Comparison of Two Approaches for Selecting Covariance Structures in the Analysis of Repeated Measures. *Communications in Statistics—Simulation and Computation*. 1998;27(3):591-604.
- 14. Kenward MG, Roger JH. Small Sample Inference for Fixed Effects from Restricted Maximum Likelihood. *Biometrics*. 1997;53:983-997.
- 15. Health Information Portability and Accountability Act (HIPAA). Available at: https://www.hhs.gov/hipaa/for-professionals/privacy/index.html

APPENDIX A: PATIENT REPORTED OUTCOMES (STUDY QUESTIONNAIRES)



| Protocol 6435 | Johnson & Johnson Vision Care, Inc. | Confidential |
|---------------|-------------------------------------|--------------|

**Protocol 6435** 

Page 96 of 177
PRO SPECIFICATION Version 1 Final 2021-04-28

Johnson & Johnson Vision Care, Inc.

| Protocol 6435 | Johnson & Johnson Vision Care, Inc. | Confidential |
|---------------|-------------------------------------|--------------|

| Protocol 6435 | Johnson & Johnson Vision Care, Inc. | Confidential |
|---------------|-------------------------------------|--------------|



### APPENDIX B: PATIENT INSTRUCTION GUIDE

Will be provided separately.

## APPENDIX A: PACKAGE INSERT (APPROVED PRODUCT)

Not Applicable, as this study uses Investigational Products.

APPENDIX D: LENS FITTING GUIDE





## APPENDIX E: PRESBYOPIC SYMPTOMS QUESTIONNAIRE

| • |
|---|

#### APPENDIX F: OCULAR DOMINANCE


#### APPENDIX G: BINOCULAR OVER REFRACTION



#### APPENDIX H:

- DETERMINATION OF NEAR ADDITION
- NEAR logMAR VISUAL ACUITY MEASUREMENT PROCEDURE
- LENS FITTING CHARACTERISTICS
- SUBJECT REPORTED OCULAR SYMPTOMS
- DETERMINATION OF DISTANCE SPHEROCYLINDRICAL REFRACTIONS
- BIOMICROSCOPY SCALE
- KERATOMETRY
- DISTANCE AND NEAR VISUAL ACUITY EVALUATION
- TORIC FIT EVALUATION
- ETDRS DISTANCE VISUAL ACUITY MEASURMENT PROCEDURE
- VISUAL ACUITY CHART LUMINANCE AND ROOM ILLUMINATION TESTING

, DETERMINATION OF NEAR ADDITION

NEAR LOGMAR VISUAL ACUITY MEASUREMENT PROCEDURE

, LENS FITTING CHARACTERISTICS

Document Number: Revision Number: 5

, SUBJECT REPORTED OCULAR SYMPTOMS

DETERMINATION OF DISTANCE SPHEROCYLINDRICAL REFRACTIONS

**Determination of Distance Spherocylindrical Refractive Error** 

Title:

, BIOMICROSCOPY SCALE

KERATOMETRY



■ DISTANCE AND NEAR VISUAL ACUITY EVALUATION

CR-6435, v1.0

Document Number: 4
## TORIC FIT EVALUATION

**Document Type:** 

Document Number: 6



Title: Toric Fit Evaluation

Document Type:

Document Number: Revision Number: 6



DISTANCE LOGMAR VISUAL ACUITY MESAUREMENT PROCEDURE



VISUAL ACUITY CHART LUMINANCE AND ROOM ILLUMINATION TESTING

Document Number: 4

Visual Acuity Chart Luminance and Room Illumination Testing

Title:

APPENDIX I: GUIDELINES FOR COVID-19 RISK MITIGATION

#### 1.0 PURPOSE

The purpose of this document is to provide guidelines for the re-opening or initiation of clinical study sites participating in Johnson & Johnson Vision Care, Inc. (JJVCI) clinical studies during the COVID-19 pandemic.

#### 2.0 SCOPE

This document provides guidelines for Johnson & Johnson Vision Care (JJVCI) to address the potential risks from COVID-19 to study subjects, investigators, study site staff, and monitors at study sites. The guidance provided in this document is in effect from the date of approval through the date of retirement of this Work Instruction. At a minimum, this Work Instruction will be reviewed and updated on a quarterly basis, as appropriate.

NOTE: Re-opening of sites outside of the US will be evaluated on a country by country basis subject to local health authority guidance.

## 3.0 **DEFINITIONS**

American Academy of Optometry (AAO): The American Academy of Optometry is an organization of optometrists based in Orlando, Florida. Its goal is to maintain and enhance excellence in optometric practice, by both promoting research and the dissemination of knowledge. The AAO holds an annual meeting, publishes a monthly scientific journal, gives credentials to optometrists through the fellowship process and publishes position statements.

American Optometric Association (AOA): The American Optometric Association, founded in 1898, is the leading authority on quality care and an advocate for our nation's health, representing more than 44,000 Doctors of Optometry (O.D.), optometric professionals, and optometry students. Doctor of Optometry take a leading role in patient care with respect to eye and vision care, as well as general health and well-being. As primary health care providers, Doctor of Optometry have extensive, ongoing training to examine, diagnose, treat and manage ocular disorders, diseases and injuries and systemic diseases that manifest in the eye. The American Optometric Association is a federation of state, student, and armed forces optometric associations. Through these affiliations, the AOA serves members consisting of optometrists, students of optometry, paraoptometric assistants and technicians. The AOA and its affiliates work to provide the public with quality vision and eye care.

**Centers for Disease Control and Prevention (CDC):** The Centers for Disease Control and Prevention is a national public health institute in the United States. It is a United States federal agency, under the Department of Health and Human Services, and is headquartered in Atlanta, Georgia.

**COVID-19:** Current outbreak of respiratory disease caused by a novel coronavirus. The virus has been named "SARS-CoV-2" and the disease it causes has been named "Coronavirus Disease 2019" (COVID-19).

Clinical Study: Voluntary research studies conducted in people and designed to answer specific questions about the safety or effectiveness of drugs, vaccines, other therapies, or new ways of using existing treatments. May also be called clinical trials, studies, research, trials, or protocols.

Clinical Study Site: Location where a clinical study is conducted, such as a doctor's office, university, or laboratory. Clinical studies are conducted by Investigators who are individual(s) responsible for the conduct of the clinical study at a study site. If a study is conducted by a team of individuals, the Investigator is the responsible leader of the team and may be called the Principal Investigator.

**Clinical Operations Manager (COM):** The Johnson & Johnson Vision Care (JJVCI) individual responsible for the overall management of a clinical trial.

| Title: | <b>Guidelines for COVID-19 Risk Mitigation</b> | |
|---|---|---|
| <b>Document Type:</b> | | |
| <b>Document Number:</b> | | <b>Revision Number: 5</b> |

**Monitor:** An individual designated to oversee the progress of a clinical study and ensure that it is conducted, recorded, and reported in accordance with the protocol, Standard Operating Procedures (SOPs), Good Clinical Practice (GCP), and applicable regulatory requirements.

**Medical Safety Officer (MSO):** Physician who has primary accountability in their product portfolio for product health and safety, and who serves as an independent medical voice for patient safety.

**Safety Management Team (SMT):** A cross-functional, collaborative team responsible for review, assessment and evaluation of medical safety data arising from any source throughout the product life cycle.

#### 4.0 GUIDANCE FOR STUDY DOCUMENTS

In alignment with recent health authority guidance, JJVCI is providing recommendations for study-related management in the event of disruption to the conduct of the clinical study. This guidance does not supersede any local or government requirements or the clinical judgement of the investigator to protect the health, safety and well-being of participants and site staff. If, at any time, a participant's safety is considered to be at risk, study intervention will be discontinued, and study follow-up will be conducted as outlined in the protocol.

During the COVID-19 pandemic, the additional risks listed below need to be considered for study participants and study personnel:

#### 4.1 Additional Risks Related to the COVID-19 Pandemic:

- The possible transmission of the Coronavirus infection and consequent complications, beyond the risk of adverse events due to the investigational device and/or procedures.
- The risk may be higher in an optometric clinical study because of the close contact the subject will have with health care professionals during the procedures and assessments (since the investigator must make the measurements close to the subject's face) and, in addition the need for multiple follow-up visits/exams which may expose the subject to other patients and/or healthcare professionals who might be transmitting the virus, even if they do not have symptoms.
- Potential disruptions to the study may be necessary due to current or future pandemic-related emergency restrictions, which may lead to delays in scheduled follow-up visits.
- Subjects experiencing an adverse event related to contact lens wear may receive delayed treatment due to COVID-19 restrictions. In this event, all assessments that can be conducted virtually will be completed by the investigator to determine the best course of treatment for the subject, including an unscheduled visit, up to discontinuation from the study, as appropriate.

If a study subject is found to have contracted COVID-19 during participation in a study, he/she will be discontinued from the study and followed until COVID-19 Adverse Event (AE) resolution.

To help minimize the above potential risks, JJVCI recommend reviewing/complying with local, state, and governmental guidance for COVID-19 risks.

JJVCI will provide the following study specific documents with language pertaining to COVID-19 risks:

#### 4.1.1 Informed Consent:

Will include information concerning the study-associated risks related to the COVID-19 pandemic in bold font and/or boxed on the first page of the Informed Consent document:

| 11110. | Guidelines for COVID-17 Risk Wingation | |
|---|---|---|
| <b>Document Type:</b> | | |
| Document Number | | Revision Number: 5 |

#### STUDY ASSOCIATED RISKS RELATED TO COVID-19 (CORONAVIRUS) PANDEMIC

Cuidolines for COVID 10 Disk Mitigation

It is important to note that this study will be conducted, at least in part, during the COVID-19 pandemic. As such, additional risks associated with the infection with COVID-19 exist for you. This is particularly important for this study due, in part, to the closeness of the doctor during the study examinations.

The potential effects of the disease are not fully known, at this time, and may include long-term serious health consequences. In severe cases, this may result in hospitalization and/or death. Based on current knowledge from the Centers for Disease Control and Prevention (CDC), those at high-risk for severe illness from COVID-19 include older adults and people with underlying medical conditions.

During this study, all appropriate measures will be taken to minimize risks including the use of personal protective equipment such as masks and gloves, as well as proper sanitization. This is in conformance to guidance from the CDC, local health departments, and the state and county in which the study doctor's office is located. However, these measures may not completely eliminate the risks associated with contracting COVID-19.

If you are found to have contracted COVID-19 or feel ill with flu-like symptoms during participation in the study, you will not be permitted to continue in-office study follow-up visits, but you will receive instructions and your condition will be monitored by the doctor and/or study staff.

#### 4.1.2 COVID-19 Risk Control Checklist (Attachment-B):

Title.

Will include COVID-19 risk control methods that are required by a site to conduct JJVCI clinical studies. The risk controls are consistent with CDC, AOA, AAO Guidance. The Principal Investigator will review/sign the study specific checklist prior to the Site Initiation Meeting.

## 4.1.3 Protocol Compliance Investigator(s) Signature Page:

Will include a statement indicating that the Principal Investigator (PI) agrees to conduct the study in compliance with all local, state, and governmental guidance's for COVID-19 risk mitigation.

I have read the suggested guidance provided by JJVCI pertaining to the COVID-19 risk mitigation, (COVID-19 Work Instruction in the Appendix of this protocol). I agree to conduct this study in compliance with local, state, governmental guidance for COVID-19 risks.

## 4.1.4 Study Site Initiation Training Slides:

Will include suggestions to help mitigate potential transmission of COVID-19. Suggestions may include maintaining social distancing in the clinical site by staggered scheduling of study patients, wearing proper PPEs, frequent disinfection, and installing shields on the slit lamp and other applicable equipment.

#### 5.0 GUIDANCE FOR REMOTE SUBJECT VISITS

Potential disruptions to the study may be necessary due to current or future pandemic-related emergency restrictions. Possible disruption of the study as a result of COVID-19 control measures may lead to delays in scheduled follow-up visits.

Subjects may be delayed in being seen for study follow up visit(s), for example due to COVID-19 control measures or due to the subject's concerns or fears about COVID-19 risk. When appropriate, the remote assessment will be conducted to the extent possible. Discussions with the subject during remote assessments may include:

Title:

Document Type:

Document Number: 5

| Procedure | Details |
|---|---|
| Subject Reported Ocular<br>Symptoms | Subjects will respond to a verbal open-ended symptoms questionnaire regarding the test article when applicable and feasible. |
| Change of Medical History<br>(Adverse Events) and<br>Concomitant Medications /<br>Therapies Review | Record any adverse events or medical history changes from the previous study visit with the subject/parents. Review the subject's concomitant medications/therapies and record any changes from the previous study visit. |
| Wearing Time and<br>Compliance | Record the average wearing time (including number of hours per day during weekdays and weekends, and number of days per week). Confirm compliance with the prescribed wear schedule. Record and discuss the lens wear compliance based on the subject's self-report. For example, the subjects will be asked the time of the day the subject typically puts on the study lenses in the morning and takes off in the evening, the number of days per week lenses were worn, and the number of consecutive days the subject didn't wear the study lenses, etc. |

The discussion with the subject will be documented in EDC under Tele-Visit and a minor protocol deviation will be noted. If during the telephone consultation, a subject states he/she wishes to discontinue participating in the study, instruct the subject to stop wearing the study lenses and schedule the subject to return to the clinic for a Final Evaluation at the at earliest possible time. Subjects should return all unused lenses to the clinic at the last visit.

Changes in study visit schedules, missed visits, or participant discontinuations may lead to missing data, including data related to protocol-specified procedures. Case report forms should capture specific information regarding the basis of missing data, including the relationship to the COVID-19 pandemic.

#### 6.0 STUDY CONDUCT DURING PANDEMIC

It is recognized that the Coronavirus Disease 2019 (COVID-19) pandemic may have an impact on the conduct of this clinical study due to, for example, self-isolation/quarantine by participants and study-site personnel; travel restrictions/limited access to public places, including Optometry Clinics; and changes in clinic procedures required to address the COVID-19 challenge.

Every effort should be made to adhere to protocol-specified assessments for study participants, including follow-up. However, if scheduled visits cannot be conducted in person at the study site it is suggested that assessments be performed to the extent possible remotely/virtually or delayed until such time that on-site visits can be resumed in order to continue participant monitoring in accordance with the protocol where possible. At each contact, participants will be interviewed to collect safety data. Key efficacy endpoint assessments should be performed if required and as feasible.

Modifications to protocol-required assessments may be permitted via COVID-19 Appendix after consultation with the participant, investigator, and the sponsor. Missed assessments/visits will be captured in the clinical trial management system for protocol deviations. Interruptions of test article wear or discontinuations of study interventions and withdrawal from the study should be documented with the prefix "COVID-19-related" in the case report form (CRF).

| Title: | Guidelines for COVID-19 Risk Mitigation | |
|---|---|---|
| <b>Document Type:</b> | | |
| <b>Document Number:</b> | | <b>Revision Number: 5</b> |

The sponsor will continue to monitor the conduct and progress of the clinical study, and any changes will be communicated to the sites and to the health authorities according to local guidance.

If a participant has tested positive for COVID-19, the investigator should contact the sponsor's responsible medical monitor to discuss initial plans for study intervention and follow-up. The medical monitor will notify the Safety Management Team of any subject(s) that have reported "COVID-19", "Asymptomatic COVID-19", or "Suspected COVID-19" adverse events within 24 hours of the notification.

Modifications made to the study conduct as a result of the COVID-19 pandemic will be summarized in the clinical study report.

COVID-19 screening procedures that may be mandated by local healthcare systems do not need to be reported as an amendment to the protocol even if done during clinical study visits.

## 6.1 Monitoring Visits

When on-site monitoring by the sponsor is not feasible, the sponsor's site monitor will contact the study site to schedule remote visits. In such cases, on-site monitoring visits will resume when feasible, with increased frequency to address the source data verification backlog.

Even with staffing limitations during this COVID-19 pandemic, all routine operations related to clinical trials should be well-documented and archived as part of standard process. When conditions permit, all parties involved in this clinical trial should communicate relevant information in a timely manner so that all relevant parties remain sufficiently informed.

## 6.1.1 Study Site Initiation:

During the period that this Work Instruction is in effect, Site Initiation Meetings and training of study site staff will be conducted remotely. The JJVCI study team will conduct training via Skype, Zoom, Microsoft Teams or similar software as well as utilize online training materials, as applicable. Study site training will be documented utilizing Site Initiation Report

On-site visits may be considered when, for example, hands-on training or evaluation of site facilities is required. While on site, the Clinical Research Associate (CRA) will follow all local, state, and governmental policies for COVID-19 Risk Mitigation, including social distancing, wearing of PPE, etc. as applicable for the location of the study site.

## 6.1.2 Interim Monitoring Visits (if applicable):

During the period that this Work Instruction is in effect, Interim Monitoring On-site visits will be kept to a minimum and include only those tasks that the CRA cannot perform remotely (e.g., source document verification, test article reconciliation, etc.).

To ensure data integrity during the conduct of all JJVC studies, clinical study teams will follow the study specific Clinical Monitoring Plan

While on site, the CRA will follow all local, state, and governmental policies for COVID-19 Risk Mitigation, including social distancing, wearing of PPE, etc. as applicable for the location of the study site.

| Title: | Guidelines for COVID-19 Risk Mitigation | Guidelines for COVID-19 Risk Mitigation |
|---|---|---|
| <b>Document Type:</b> | | |
| <b>Document Number:</b> | | <b>Revision Number: 5</b> |

## 6.1.3 Study Site Closure:

During the period that this Work Instruction is in effect, the duration of the Study Site Closure Visit will be limited to tasks that the CRA cannot perform remotely (e.g., source document verification, test article final reconciliation and return, etc.).

| 1 lue: | Guidelines for COVID-19 Risk Willigation | |
|---|---|---|
| <b>Document Type:</b> | | |
| <b>Document Number:</b> | | <b>Revision Number: 5</b> |

### **Attachment A: Study Site Correspondence**

XXXX XX, 2020

## Re: COVID-19 Mitigation Plan, << CR-xxxx/protocol title>>

Dear << Principal Investigator>> and Study Team,

Coronavirus (COVID-19) has impacted several communities and business activities over the past several months. While we work toward the successful conduct of clinical studies, our commitment continues to be the safety of patients, healthcare professionals, and to our communities.

Therefore, we would like to share the following revisions/additions related to the above referenced Johnson & Johnson Vision Care company sponsored clinical trial(s) you are currently working on or considering participation within.

#### **Protocol:**

Guidelines for COVID-19 Risk Mitigation provided in the Appendix section.

#### **Protocol Signature Page:**

 Will include a statement indicating the Principal Investigator agrees to conduct the study in compliance with all local, state, and governmental guidelines for COVID-19 risk mitigation.

## **Informed Consent:**

• Will include information concerning the study-associated risks related to the COVID-19 pandemic in bold font and/or boxed on the first page of the Informed consent document.

## **COVID-19 Risk Control Checklist for Clinical Studies:**

• Will include COVID-19 risk control measures that are required to ensure the safety and health of subjects, site staff and monitors during the pandemic.

We want to encourage the need for open lines of communication about potential challenges you may foresee as the result of the current COVID-19 situation. Therefore, we encourage you to regularly connect with your respective Johnson & Johnson clinical study team (Clinical Research Associate (CRA), Lead CRA or Study Managers).

Thank you for your continued engagement, collaboration, and dedication to your study subjects during this challenging time.

Please file this letter in your site file study correspondence.

| Title: | Guidelines for COVID-19 Risk Mitigation | |
|---|---|---|
| <b>Document Type:</b> | | |
| <b>Document Number:</b> | | <b>Revision Number: 5</b> |

## **COVID-19 Risk Control Checklist (Attachment-B):**

Study Number Site Number Principal Investigator (PI) Name

The following COVID-19 risk control methods are required to conduct Johnson & Johnson Vison Care clinical studies. Please review the following requirements and Initial each requirement.

| PI Initials | General Site Safety Planning Measures |
|---|---|
| | Signage within site describing Risk Control methods |
| | Social Distancing practices throughout site (waiting rooms, lobby, exam rooms, etc.) |
| | Non-contact thermometer available to assess temperatures of staff and patients |
| | Training on patient flow and physical distancing in waiting room |
| | Establish longer time frame between patient appointments to reduce persons in the site |
| | Staff should receive job-specific training on PPE and demonstrate competency with selection and proper use of PPE and wear at all times during interactions with subjects (e.g., putting on and removing without self-contamination) |

| PI Initials | Site Staff Daily Safety Measures |
|---|---|
| | As part of routine practice, site staff should regularly monitor themselves for fever and symptoms |
| | of COVID-19, including temperature checks |
| | Any staff member (including non-study clinic staff and Investigators) showing signs of being sick |
| | or testing positive for COVID-19 must not be permitted to work on activity that may expose study |
| | related staff and subject and the Sponsor shall be informed |
| | NOTE: Inform JJVC in 24 hours of any COVID-19 cases and all potential exposure during |
| | the clinical study. |
| | Ensure that all staff wear a mask |
| | Gloves should be required when working directly with patients and changed between each patient |
| | Have staff thoroughly wash hands for at least 20 seconds or use an alcohol-based hand sanitizer |
| | when they arrive, before and after each patient, before eating and after using the bathroom. |
| | Cleaning and disinfection procedures for exam rooms and instruments or equipment between |
| | patients with gloves. |
| | Cleaning and disinfection procedures for commonly touched surfaces (doors, chairs, computers, |
| | phones, etc.) with gloves. |

| PI Initials | Before a Patient or Study Visit: |
|---|---|
| | Patients should be asked prior to entering the site about fever and respiratory illness and whether they or a family member have had contact with another person with confirmed COVID-19 in the past 14 days. Patients exhibiting signs of being sick should be rescheduled when their symptoms resolve. |
| | Instruct patients that companions should remain outside of the facility and not accompany the patient into the facility unless they are a parent/guardian of the patient or if they are a true caregiver and need to assist the patient |
| | Request the patient to call or text the office upon arrival so entrance to and movement through facility can be coordinated by site staff |

| Document Type: | |
|-------------------------|--------------------|
| <b>Document Number:</b> | Revision Number: 5 |

| PI Initials | Patients Entering the site: |
|---|---|
| | Temperature checks utilizing a non-contact thermometer for all patients and companions entering |
| | the site. |
| | All patients and companions must wear cloth or disposable mask at all times in the site |
| | Maintain social distancing. Waiting rooms or lobbies should be as empty as possible. Advise |
| | seated patients to remain at least 6 feet from one another. |
| | Communal objects in (e.g. toys, reading materials, etc.) should be removed or cleaned regularly. |

I certify that I have read and agree to implement all the listed COVID-19 Risk Control Measures required for the conduct of Johnson & Johnson Vision Care studies.

Principal Investigator Signature and Date

| Title: | <b>Guidelines for COVID-19 Risk Mitigation</b> | |
|---|---|---|
| <b>Document Type:</b> | | |
| <b>Document Number:</b> | | Revision Number: 5 |

Suidelines for COVID 10 Disk Mitigation

#### RESOURCE LINKS

#### **US Resource Links**

**OSHA** Training

https://www.osha.gov/SLTC/covid-19/controlprevention.html

Personal Protective Equipment (PPE) Training

CDC: https://www.cdc.gov/coronavirus/2019-ncov/hcp/using-ppe.html

I&R Training

ACUVUE® LensAssist: <a href="https://www.acuvue.com/lensassist">https://www.acuvue.com/lensassist</a>

Clinic Preparedness Guides

CDC: https://www.cdc.gov/coronavirus/2019-ncov/hcp/clinic-preparedness.html AOA: https://aoa.uberflip.com/i/1240437-aoa-guidance-for-re-opening-practices-covid-19/1?m4= American Optometric Association: https://www.aoa.org/optometry-practice-reactivation-preparednessguide

In-Office Disinfection of Multi-Patient Use Diagnostic Contact Lenses https://www.gpli.info/wp-content/uploads/2020/03/2020-01-15-in-office-disinfecting-of-diagnosticlenses.pdf

## **OUS Resource Links**

- Updates on local regulations in Hong Kong https://www.coronavirus.gov.hk/eng/index.html
- Resumption of optical services in England: Letter from Matt Neligan and Poonam Sharma https://www.england.nhs.uk/coronavirus/wp-content/uploads/sites/52/2020/04/C0601-reopening-of-opticalservices-letter-17-june-2020.pdf
- NHS Optical Letter https://www.england.nhs.uk/coronavirus/wp-content/uploads/sites/52/2020/04/C0127-optical-letter-1-april-2020.pdf
- The College of Optometrists primary eye care COVID-19 guidance: Red phase https://www.college-optometrists.org/the-college/media-hub/news-listing/coronavirus-covid-19-guidancefor-optometrists.html
- The College of Optometrists COVID-19: College updates https://www.college-optometrists.org/the-college/media-hub/news-listing/coronavirus-2019-advice-foroptometrists.html#CollegeGuidelines
- Infection Control Guidelines. (n.d.). Retrieved from Canadian Association Of Optometrists: https://opto.ca/sites/default/files/resources/documents/infection control guidelines 2016.pdf
- Infection prevention and control for COVID-19: Interim guidance for outpatient and ambulatory care settings. (2020, May 23 May). Retrieved from Government of Canada: https://www.canada.ca/en/publichealth/services/diseases/2019-novel-coronavirus-infection/guidance-documents/interim-guidanceoutpatient-ambulatory-care-settings.html

| Title: | Guidelines for COVID-19 Risk Mitigation | |
|---|---|---|
| <b>Document Type:</b> | | |
| <b>Document Number:</b> | | <b>Revision Number: 5</b> |

- Information for Members On Coronavirus (COVID-19). (n.d.). Retrieved from Canadian Association Of Optometrists:
  - https://opto.ca/sites/default/files/resources/documents/information\_for\_members\_on\_coronavirus.pdf
- Coronavirus (COVID-19) resources for health professionals, including aged care providers, pathology providers and health care managers. (2020, September 24). Retrieved from Australian Government Department of Health:
  - https://www.health.gov.au/resources/collections/coronavirus-covid-19-resources-for-health-professionals-including-aged-care-providers-pathology-providers-and-health-care-managers
- Environmental Cleaning and Disinfection Principles for COVID-19. (n.d.). Retrieved from Australian Government Department of Health: https://www.health.gov.au/sites/default/files/documents/2020/03/environmental-cleaning-and-disinfection-principles-for-covid-19.pdf
- Infection control guidelines and advice. (n.d.). Retrieved from Optometry Australia: https://www.optometry.org.au/practice-professional-support/coronavirus-covid-19-what-optometrists-need-to-know/covid-19-clinical-advice/infection-control-guidelines-and-advice/

## PROTOCOL COMPLIANCE INVESTIGATOR(S) SIGNATURE PAGE

Protocol Number and Title: CR-6435 Evaluation of Daily Disposable Silicone Hydrogel Multifocal Toric Contact Lenses

Version and Date: 1.0, 12 May 2021

I have read and understand the protocol specified above and agree on its content.

I agree to conduct this study according to ISO 14155, GCP and ICH guidelines, the Declaration of Helsinki, United States (US) Code of Federal Regulations (CFR), and the pertinent individual country laws/regulations and to comply with its obligations, subject to ethical and safety considerations. The Principal Investigator is responsible for ensuring that all clinical site personnel, including Sub-Investigators adhere to all ICH<sup>2</sup> regulations and GCP guidelines regarding clinical trials during and after study completion.

I will assure that no deviation from or changes to the protocol will take place without prior agreement from the Sponsor and documented approval from the Institutional Review Board (IRB), except where necessary to eliminate an immediate hazard(s) to the trial participants.

I am responsible for ensuring that all clinical site personnel including Sub-Investigators adhere to all ICH<sup>2</sup> regulations and GCP guidelines regarding clinical trials during and after study completion.

All clinical site personnel involved in the conduct of this study have completed Human Subjects Protection Training.

I agree to ensure that all clinical site personnel involved in the conduct of this study are informed about their obligations in meeting the above commitments.

I shall not disclose the information contained in this protocol or any results obtained from this study without written authorization.

I have read the suggested guidance provided by JJVCI pertaining to the COVID-19 risk mitigation, (COVID-19 Work Instruction in the Appendix I of this protocol). I agree to conduct this study in compliance with local, state, governmental guidance for COVID-19 risks.

| Principal Investigator: | | |
|-------------------------|------------------------------------------|------|
| | Signature | Date |
| | Name and Professional Position (Printed) | _ |
| Institution/Site: | | |
| | Institution/Site Name | |
| | Institution/Site Address | |